# **Clinical Study Protocol**

NRX101-003

## Study Title: A Randomized, Double-Blind Controlled Comparison of NRX-101 to Lurasidone for Adults with Bipolar Depression and Subacute Suicidal Ideation or Behavior

Principal Investigator Andrew Nierenberg, MD

Study Sponsor NRx Pharma, Inc., Inc.

1201 N Market Street; Suite 111

Wilmington, DE 19801

IND Number 129194

Phase 2b

Document Status Final

Version, Date 4.0 09NOV2023

This document is the confidential property of NRx Pharmaceuticals, Inc. and may not be disclosed or used without the prior written consent of NRx Pharmaceuticals, Inc.

NRX-101 003  09 NOVEMBER 2023

### 1. CONTACT INFORMATION

| Role in Study | Name | Telephone |
|-------------------------------|-----------------------------|--------------|
| NeuroRx, Inc. Chief Scientist | Jonathan C. Javitt, MD, MPH | 202-340-1352 |
| NeuroRx, Inc. Medical Monitor | Martin Brecher, MD | 215-208-8580 |
| Principal Investigator | Andrew Nierenberg, MD | 617-724-0837 |

## 2. Study Synopsis

| Name of<br>Investigational<br>Product: | NRX-101 |
|---|---|
| Name of Active<br>Ingredient: | NRX-101: Oral capsule containing a fixed-dose combination of D-cycloserine (DCS) + lurasidone HCl (NRX-101) |
| Reference<br>Product(s): | Lurasidone HCl ("lurasidone") + placebo |
| Title of Study: | A Randomized, Double-Blind, Controlled Comparison of NRX-101 to lurasidone for Treatment of Bipolar Depression in Adults with Subacute Suicidal Ideation or Behavior |
| Short Title: | Comparison of NRX-101 to Standard of Care for Bipolar Depression with Subacute Suicidal Ideation or Behavior |
| Phase of Development: | Phase 2b |
| Study Sites: | 10-20 sites located in the United States |
| Total Patient<br>Number: | 74 participants |
| Study Duration: | Up to 10-weeks per patient: Screening 1 up to 10 days, Treatment from Day 1 to Day 42, and Follow-up on Day 70 |
| Background and<br>Rationale: | There is no currently-approved pharmacotherapy for patients with Severe Bipolar Depression and Suicidal Ideation or behavior. The purpose of this phase 2b trial is to determine whether patients with Severe Bipolar Depression and subacute Suicidal Ideation or Behavior (i.e. those not requiring inpatient care) can be treated effectively with NRX-101. |
| Objectives: | <ul> <li>Primary Objective:</li> <li>To test the hypothesis that treatment with NRX-101 is superior to lurasidone (a standard of care medicine) in improving symptoms of depression as measured by the Montgomery Åsberg Depression Rating Scale (MADRS-10) total score in adults with severe bipolar depression and subacute suicidal ideation or behavior (SSIB).</li> <li>Key Secondary Objectives:</li> <li>To test the hypothesis that NRX-101 is superior to lurasidone in reducing suicidal ideation or behavior as measured by the Clinical Global Impression of Severity of Suicidality Scale (CGI-SS).</li> <li>To test the hypothesis that NRX-101 is superior to lurasidone in time to treatment failure as defined as: study discontinuation due to adverse events; psychiatric hospitalization; or requiring a change in antidepressant treatment.</li> </ul> |

#### Additional Secondary Objectives:

- To test the hypothesis that treatment with NRX-101 is superior to standard of care (lurasidone) in reducing suicidal ideation (MADRS item 10).
- To test the hypothesis that treatment with NRX-101 is superior to lurasidone in reducing the frequency of suicidal thoughts, suicidality and risk (SIBAT Module 7).
- To test the hypothesis that treatment with NRX-101 is superior to treatment with lurasidone in the subgroup of participants recently (i.e. within two weeks of enrollment) treated with approved medications for bipolar depression (olanzapine/fluoxetine, quetiapine, cariprazine, lumateprone, or lurasidone).

#### Safety Objectives:

- To test the hypothesis that treatment with NRX-101 is superior to lurasidone (a standard of care drug) in reducing suicidality in depressed bipolar patients with SSIB, as measured by the Columbia Suicide Severity Rating Scale (C-SSRS).
- To test the hypothesis that participants treated with NRX-101 are less likely to suffer from akathisia than those treated with lurasidone as measured by the Barnes Akathisia Rating Scale (BARS).
- To test the hypothesis that fewer participants treated with NRX-101 will be discontinued for lack of efficacy or exacerbation of suicidality than participants treated with lurasidone.

# **Efficacy Endpoint(s):**

#### Primary Endpoint:

• Change from baseline over 42 days in MADRS total score.

#### **Key Secondary Endpoints:**

- Change from baseline over 42 days in CGI-SS.
- Time to treatment failure in each arm.

#### Additional Secondary Endpoints:

- Mean change from baseline in Suicidal Thoughts on the MADRS (MADRS item 10).
- Change from baseline to Day 14 in MADRS total score.
- Change from baseline in each item of the Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 (clinical global impressions of frequency of suicidal thinking, severity of suicidality, and imminent and long-term risks).
- Change from baseline to endpoint (Day 42/exit) in MADRS total score in the subgroup of participants who were recently (within 2-weeks) on approved medications for bipolar depression.
- Percent in remission from suicidality at Day 42/exit (exploratory endpoint).

#### **Study Design:**

A multicenter, randomized, stratified, double-blind, parallel-group, two-arm outpatient study of 74 participants comparing NRX-101 to lurasidone in a 1:1 ratio for the treatment of bipolar depression in participants with Subacute Suicidal Ideation or behavior and not requiring hospitalization, as reflected by a

rating of 3 or 4 on the C-SSRS at screening. A priori sample size suggests > 90% power based on effect size of >1 seen in phase 2 STABIL-B trial. There is 80% power to detect a 0.66 effect size; a 0.462 effect size would reach two-sided p=0.05.

Two interim analyses are planned. The first interim analysis (IA) assessing safety will be conducted six weeks after the first 30-35 participants have been followed for 6 weeks and the second IA assessing futility (primary efficacy endpoint) will be performed after the first 45-50 participants have been followed for 6 weeks.

Each interim analysis has a different objective with neither interim analysis spending any Type 1 error. The study will be stopped at the first interim analysis if Serious Adverse Events are deemed statistically significantly more common in the NRX-101 group compared to the lurasidone group in a manner deemed by the DMC to pose a potential danger to human subjects. The study will be stopped at the second IA for futility if the conditional power (CP) is less than 10%. In the event that the study is not stopped for either safety or futility, then enrollment will continue until a total of 74 subjects are randomized. This preserves two-sided p=0.05 for the final analysis.

#### **Inclusion Criteria:**

A patient is eligible for inclusion in this study only if all of the following criteria apply:

- 1. 18 to 65 years of age, inclusive, at Screening.
- 2. Able to understand and provide written and dated informed consent prior to Screening.
- 3. Deemed likely to comply with the study protocol, including communication of adverse events (AEs) and other clinically important information, including adherence to the text messaging component of the trial.
- 4. Will follow medical directions for psychiatric care, as appropriate, per the standard of care.
- 5. Resides in a stable living situation. A stable living situation will be defined as a minimum of 3 months at the same address with a reasonable expectation that the situation will continue such that the patient's ability to participate in the study will not be affected. Please note that housing in a shelter of any kind will not be deemed stable housing.
- 6. Previously diagnosed and treated for Bipolar Disorder (BD) I or II according to the criteria defined in the DSM-V.
- 7. Has an identified reliable informant/care partner that is willing to provide information and/or supportive care as necessary.
- 8. The diagnosis of BD will have been made by a psychiatrist or other qualified licensed psychiatric provider able to render a diagnosis and be supported by the MINI 7.0.2.
- 9. Treatment with a medication indicated for use in bipolar disorder in the past five years (See Appendix 4 for list).

- 10. Confirmed active suicidal ideation, (without the intention to act) as evidenced by an answer of 'Yes' on item 3 and/or item 4 and not requiring hospitalization at Screening and an answer of "No" on item 5 of the C-SSRS within 4-weeks of Screening.
- 11. A total score greater than or equal to 30 on the 10 items of the MADRS.
- 12. No co-morbidities as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and electrocardiogram (ECG) which might interfere with compliance or the ability to assess efficacy or safety.
- 13. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following criteria, and agrees to continue use of the same method of birth control for the duration of study participation:
  - a. Non-childbearing potential: physiologically incapable of becoming pregnant (i.e., permanently sterilized [status post-hysterectomy, bilateral tubal ligation], or post-menopausal with last menses at least one year prior to Screening); or
  - b. Childbearing potential, and meets the following criteria:
    - i. Use of any form of hormonal birth control for at least 2 months prior to Screening, on hormone replacement therapy that started prior to 12 months of amenorrhea, using an intrauterine device (IUD) for at least 1 month prior to Screening, in a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.
    - ii. Negative urinary pregnancy test at Screening, confirmed by a second negative urinary pregnancy test at Day 1, prior to receiving study treatment.
- 14. Body mass index (BMI) between 18-40 kg/m<sup>2</sup>; BMI up to 45 kg/m<sup>2</sup> is allowed with Medical Monitor review and approval.
- 15. If receiving concurrent psychotherapy, the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation.
- 16. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, maximum 2 mg daily, or trazodone) will be allowed if the therapy has been stable for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
- 17. Concurrent treatment with benzodiazepines is allowed up to a maximum dose 2mg/daily used for anxiety if therapy has been stable relative to dose and schedule for at least four-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
- 18. If women are receiving hormone replacement therapy or estrogen replacement, the therapy has been stable for at least 3 months prior to screening and is expected to remain stable for the duration of the study participation.

#### **Exclusion criteria:**

A patient is ineligible for inclusion in this study if any of the following criteria apply:

- 1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
- 2. Female who is pregnant or breastfeeding.
- 3. Female with a positive pregnancy test at Screening or prior to randomization.
- **4.** Current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to Screening. (Note: Substance use disorder cannot be the precipitant for study entry).
- 5. A lifetime history of
  - a. phencyclidine (PCP)/ketamine drug abuse, or
  - b. failed use of ketamine for depression or suicidality.
- 6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
- 7. History of anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified (NOS), or other specified feeding and eating disorders (OSFED) within 3 years of Screening.
- 8. Has dementia, delirium, amnestic, or any other cognitive disorder.
- 9. Current major psychiatric disorder, diagnosed at Screening with the MINI 7.0.2 which is the primary focus of treatment, with bipolar disorder as the secondary focus of treatment, within the past 6 months.
- 10. Estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m<sup>2</sup> using the Cockcroft-Gault formula.
- 11. A clinically significant abnormality on the Screening physical examination that may affect safety or study participation, or that may confound interpretation of study results according to the study clinician.
- 12. Current episode of:
  - a. Myocardial infarction within 1 year of Screening.
  - b. Diagnosis of angina pectoris.
  - c. Prolonged QTc interval, as measured by Fridericia's correction formula (QTcF) ≥450 msec at Screening for males or ≥ 470 msec for females on 2 of 3 measurements at least 15 minutes apart prior to randomization on Day 1.
- 13. Diagnosis of chronic lung disease, excluding asthma.
- 14. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS
- 15. History of significant head trauma within the past two years.

- 16. Diabetes mellitus fulfilling any of the following criteria:
  - a. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 percent at Screening.
  - b. Admitted to the hospital for treatment of diabetes mellitus or diabetes mellitus—related illness in the past 12 weeks.
    - c. Not under physician care for diabetes mellitus.
  - d. Not on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to Screening.
  - e. Not on the same dose of oral thiazolidinediones (glitazones) for the 8 weeks prior to Screening.
- 17. Any current or past history of any physical condition which, in the opinion of the investigator, may put the patient at risk or interfere with study results interpretation.
- 18. Diagnosis of HIV/AIDS.
- 19. Diagnosis of Hepatitis C.
- 20. On exclusionary concomitant psychotropic and non-psychotropic medications (see Appendix 1).
- 21. Prescribed more than one agent in each of the following categories at randomization:
  - a. Approved SSRIs.
  - b. Approved serotonin and norepinephrine reuptake inhibitors (SNRIs).
  - c. Approved tetracyclic antidepressants (TeCAs).
- Note: Any/all 5hT2A medications will be discontinued at study entry. Participants currently on Lurasidone will be randomized to either standard of care or NRX-101 at the indicated starting dose.
- 22. Currently prescribed oxcarbazepine or carbamazepine.
- 23. Exclusionary laboratory values or any other clinically significant abnormal laboratory result at Screening. Within normal limits (WNL) will be determined based on lab values of the local lab used.
- 24. Known allergies to lurasidone or Latuda<sup>®</sup>, cycloserine or Seromycin<sup>®</sup>, or the following excipients: mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or hydroxypropylmethylcellulose (HPMC).
- 25. Participation in any clinical trial with an investigational drug or device within the past month or planned concurrent study participation.
- 26. Study site personnel and/or persons employed by NRx Pharma, Inc., the Contract Research Organization (CRO), the investigator, or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate family member (i.e., spouse, parent, child, or sibling [biological or legally adopted]) of such persons.
- 27. Positive urine toxicity screening for use of any cocaine, opiates, non-prescribed amphetamines, or non-prescribed barbiturates. (Note: cannabinoids or marijuana use is not exclusionary, unless patient meets the DSM-5 criteria for cannabis withdrawal).

| | 28. Signs and symptoms of active or residual COVID-19, or unresolved symptoms of COVID-19 that impact health, e.g. requirements for oxygen supplementation, etc. Discharged from an inpatient hospitalization for more than 48 hours for COVID-19 within the past 28 days. |
|---|---|
| Analysis Sets: | For efficacy analyses, the intent-to-treat (ITT) population is defined as all participants who are randomized and receive at least one dose of investigational product and have evaluable data from at least one subsequent visit. For safety analyses; the Safety population will include data from all participants who are randomized and receive at least one dose of investigational product. |
| Pharmacokinetic<br>Assessments: | None |
| Safety<br>Assessments: | The safety of NRX-101 will be assessed via: • Adverse Events • Vital signs (blood pressure, heart rate), weight |
| | • 12-lead ECGs |
| | Clinical laboratory evaluations |
| | Physical examination findings |
| | Other Assessments: |
| | Mean change from baseline to endpoint (Day 42/exit) in C-SSRS score |
| | Mean change from baseline to Day 14 in C-SSRS score |
| | Mean change in BARS through Day 42 to assess akathisia |
| | Rates of discontinuation between arms |
| Dosage, Route of Administration, | On Day 1, eligible participants will be randomized to blinded NRX-101 or lurasidone and placebo capsules administered twice daily (BID). |
| Investigational product will be titrated over 2 days. In the case of randomizat to NRX-101, the blinded investigational product will consist of daily doses o 700 mg DCS and 33 mg lurasidone and increasing the dose to 950 mg DCS a 66 mg lurasidone on second day. The total daily NRX-101 maintenance dose Day 3 through Day 42 is 950 mg DCS and 66 mg lurasidone. In the event a patient experiences agitation or psychosis, a blinded up-titration is permitted. Similarly, a blinded step-down titration is allowed for somnolence. In order to maintain the blind, lurasidone/placebo capsules will be administered to ensur participants take the same number of capsules with each dose administration. NRX-101 is supplied in capsules that contain 237.5 mg or 175 mg of DCS and second capsule that contains 8.25 mg, 16.5 mg, or 33 mg of lurasidone. In order to maintain the blind, lurasidone/placebo capsules will be administered to ensur participants take the same number of capsules with each dose administration. | |
| | In the case of randomization to lurasidone, the blinded investigational product will start with doses of 33 mg lurasidone and increasing the dose to 66 mg. The total daily lurasidone maintenance dose for Day 3 through Day 42 is 66 mg. |
| Endpoint<br>Adjudication | All rating sessions for MADRS-10 and C-SSRS will be recorded as audio files and reviewed by central master-raters with >25 years' experience. Any MADRS-10 total score the differs by more than three points from the master-rater score |

| | will be deemed non-congruent. All non-congruent subject-visits from any site with >10% non-congruent scores will be sent to an independent adjudicator previously determined to have >90% concordance with study master raters on standardized training data. In the event of adjudication as above, the independent outside rater score shall be considered as the subject-visit primary study endpoint. |
|---|---|
| Statistical<br>Methods: | All randomized participants will be evaluated for depression (MADRS) suicidality (C-SSRS), and other efficacy endpoints while on the study. Analyses will be conducted under ICH E9 (R1) guidelines. Change from baseline in MADRS total scores through study exit to compare treatments will be analyzed using Mixed Model Repeated Measures analysis (SAS PROC MIXED) with Last Observation Carried Forward (LOCF) containing BPI rating scale (none, any) and evidence of a suicidal event in their lifetime (none, any) as stratification factors. Additional analyses will alternatively rely on multiple imputation to assess the impact of dropouts. The NRX-101 and lurasidone treatment groups will be compared using stratified and unstratified log rank tests, as well as a proportional hazard model for time to relapse. |
| Sample Size<br>Calculation: | Participants will be randomized in a 1:1 ratio (NRX-101:lurasidone). With 37 participants per group, there is an 80 percent power to detect a mean 8.85-unit advantage for NRX-101 vs lurasidone for the CFB to Day 42, assuming a SD of 13.4 for NRX-101 versus lurasidone at 6 weeks for a two-sided hypothesis test with two-sided 5 percent Type I error. This equates to a 0.66 effect size. |
| Interim Analysis | Two interim analyses are planned. The first interim analysis (IA) assessing safety will be conducted six weeks after the first 30-35 participants have been followed for 6 weeks and the second IA assessing futility (primary efficacy endpoint) will be performed after the first 45-50 participants have reached 42 days post-randomization. Each interim analysis has a different objective with neither interim analysis spending any Type 1 error. The study will be stopped at the first interim analysis if Serious Adverse Events are deemed statistically significantly more common in the NRX-101 group compared to the lurasidone group in a manner deemed by the DMC to pose a potential danger to human subjects. The study will be stopped at the second IA for futility if the conditional power (CP) is less than 10%. In the event that the study is not stopped for either safety or futility, then enrollment will continue until a total of 74 subjects are randomized. This preserves two-sided p=0.05 for the final analysis. |

#### 3. PROTOCOL SIGNATURE PAGE

I have read this protocol and agree to adhere to the requirements. I will provide copies of this protocol and all pertinent information to the study personnel under my supervision. I will discuss this material with them and ensure they are fully informed regarding the conduct of the study according to 21 Code of Federal Regulations (CFR) parts 50, 54, 56 and 812, 45 CFR 46, to Good Clinical Practice (GCP), as described in International Conference on Harmonisation (ICH) guidelines E6 and E, and to Institutional Review Boards.

| Clinical Site Investigator Signature | Date |
|------------------------------------------------|------|
| Clinical Site Investigator Printed Name | |
| Sponsor Signature | |
| Jonathan C. Javitt, MD, MPH<br>Chief Scientist | |
| Sponsor Signature | - |
| Andrew Nirenberg, MD | |
| Principal Investigator | |

NRX-101 003  09 NOVEMBER 2023

## 4. TABLE OF CONTENTS

| C | OVE | R PAGE | 1 |
|----|-------|----------------------------------------------------|----|
| 1. | CO | ONTACT INFORMATION | 2 |
| 2. | ST | TUDY SYNOPSIS | 3 |
| 3. | | ROTOCOL SIGNATURE PAGE | |
| 4. | TA | ABLE OF CONTENTS | |
| | 4.1 | List of Tables | 15 |
| | 4.2 | List of Figures | 15 |
| 5. | | BBREVIATIONS | |
| 6. | IN | TRODUCTION | |
| | 6.1 | Suicidal Ideation and Behavior in Bipolar Disorder | |
| | 6.2 | Current Treatment Options | 18 |
| | 6.3 | Preclinical Models of Anxiety and Akathisia | 19 |
| | 6.4 | Clinical Experience with DCS | 19 |
| | 6.5 | Investigational Therapy | 21 |
| | 6.6 | Dose Selection | 21 |
| 7. | OI | BJECTIVES | 22 |
| | 7.1 | Primary Objective | 22 |
| | 7.2 | Key Secondary Objectives. | 22 |
| | 7.3 | Additional Secondary Objectives | 22 |
| | 7.4 | Safety Objectives | 23 |
| | 7.5 | Overview | 23 |
| 8. | SE | ELECTION OF PARTICIPANTS | 24 |
| | 8.1 | Inclusion Criteria | 24 |
| | 8.2 | Exclusion Criteria | 25 |
| 9. | ST | TUDY VISITS | 28 |
| | 9.1 | Study Visits | 28 |
| | 9.1 | 1.1 Screening Period | 30 |
| | 9.1 | 1.2 Treatment and Follow-up Periods | 30 |
| | 9.1 | 1.3 Early Termination Visit | 31 |
| 1( | ). TF | REATMENT OF PARTICIPANTS | 31 |
| | 10.1 | Investigational Drug Dose and Administration | 31 |
| | 10.2 | Investigational Product | 31 |

| 10.3 Investigational Product Titration | 32 |
|---|---|
| 11. INVESTIGATIONAL PRODUCT MATERIALS AND MANAGEMENT | 33 |
| 11.1 Packaging and Labeling | 33 |
| 11.1.1 Storage | 35 |
| 11.1.2 Accountability | 35 |
| 11.1.3 Handling and Disposal | 35 |
| 11.2 Study Drug Monitoring | 35 |
| 12. EFFICACY ASSESSMENTS | 35 |
| 12.1 Montgomery Asberg Depression Rating Scale (MADRS) | 35 |
| 12.2 Clinical Global Impression-Severity for Suicide | 36 |
| 12.3 Brief Psychiatric Rating Scale (BPRS psychosis subscale) | 36 |
| 12.4 Concise Health Risk Tracking – Self Report (CHRT-SR) and Clinician Rating (CHRT-C) | 36 |
| 13. OTHER DIAGNOSTIC INSTRUMENTS | 36 |
| 13.1 Mini International Neuropsychiatric Interview (MINI) 7.0.2 | 36 |
| 13.2 Bipolarity Index (BPI) | 36 |
| 14. ASSESSMENT OF EFFICACY | 37 |
| 14.1 Primary Efficacy Endpoint | 37 |
| 14.2 Key Secondary Efficacy Endpoints | 37 |
| 14.3 Additional secondary efficacy endpoints: | 37 |
| 15. ASSESSMENT OF SAFETY | 37 |
| 15.1 Safety Scales | 37 |
| 15.1.1 Columbia Suicide Severity Rating Scale (C-SSRS) | 37 |
| 15.1.2 Patient Rated Inventory of Side Effects (PRISE) | 38 |
| 15.1.3 Barnes Akathisia Scale (BARS) | 38 |
| 15.2 Adverse Events and Serious Adverse Events | 38 |
| 15.2.1 Definition of Adverse Events | 38 |
| 15.2.2 Adverse Event Intensity and Relationship | 39 |
| 15.2.3 Recording of Adverse Events | 40 |
| 15.2.4 Definition of Serious Adverse Events | 40 |
| 15.2.5 Reporting Serious Adverse Events | 41 |
| 15.2.6 Anticipated Serious Adverse Events | 41 |
| 15.3 Concomitant Medications, Therapies, and Alcohol Restrictions | 42 |

| 15.3.1 Concomitant Medications | 42 |
|------------------------------------------------------------------|----|
| 15.3.2 Concomitant Therapy | 43 |
| 15.3.3 Alcohol Restrictions | 43 |
| 15.3.4 Positive Drug Screen | 43 |
| 15.4 Laboratory/Diagnostic Procedures | 44 |
| 15.5 Physical Examinations, Vital Signs, Height, and Weight | 44 |
| 15.6 Electrocardiograms | 44 |
| 15.7 Study Monitoring by the Drug Safety Monitoring Board (DSMB) | 44 |
| 16. STATISTICS | 45 |
| 16.1 Randomization | 45 |
| 16.2 Study Populations | 45 |
| 16.3 Hypothesis Tests | 45 |
| 16.3.1 Treatment Comparisons | 45 |
| 16.3.2 Primary Hypothesis | 45 |
| 16.3.3 Key Secondary Hypotheses | 46 |
| 16.4 Efficacy Endpoints | 47 |
| 16.4.1 Primary Efficacy Endpoints | 47 |
| 16.4.2 Secondary Efficacy Endpoints | 47 |
| 16.4.3 Other Exploratory Efficacy Endpoints | 47 |
| 16.4.4 Other Efficacy Endpoints of Interest | 48 |
| 16.4.5 Diagnostic Metric | 48 |
| 16.5 Safety Assessments | 48 |
| 16.5.1 Overall Adverse Events | 48 |
| 16.5.2 Other Safety Measures | 49 |
| 16.6 Sample Size Calculations | 49 |
| 16.6.1 Background | 49 |
| 16.6.2 Power and Significance | 49 |
| 16.6.3 Interim Analyses | 50 |
| 16.7 Adjudication of Primary Endpoint | 50 |
| 16.8 Statistical Analysis Approach | 51 |
| 16.8.1 Software | 51 |
| 16.8.2 Display Formats | 51 |
| 16.8.3 Conventions | 51 |

| 16.8. | 4 Estimand Structure | 51 |
|---|---|---|
| 16.8. | 5 General Methodology | 53 |
| 16.8. | 6 Other Time to Event Efficacy Endpoints | 53 |
| 16.8. | 7 Secondary Efficacy Endpoints | 54 |
| 16.8. | 8 Other Endpoints of Interest | 54 |
| 16.8. | 9 Safety Endpoints | 55 |
| 17. DIRI | ECT ACCESS TO SOURCE DATA/DOCUMENTS | 55 |
| 17.1 S | tudy Monitoring | 55 |
| 17.2 A | udits and Inspections | 57 |
| 17.3 Ir | nstitutional Review Board (IRB) | 57 |
| 18. QUA | LITY CONTROL AND QUALITY ASSURANCE | 57 |
| 18.1 S | ource Data and Records | 57 |
| 18.2 R | eporting Study Data | 58 |
| 18.2. | 1 Clinical Trial Registry | 58 |
| 18.3 C | onfidentiality of Patient Data | 58 |
| 19. ETH | ICAL CONSIDERATIONS | 59 |
| 19.1 E | thical Conduct of the Study | 59 |
| 19.2 P | atient Information and Consent | 59 |
| 20. REF | ERENCES | 60 |
| 21. APP | ENDICES | 63 |
| 4.1 List | t of Tables | |
| Table 1 | Schedule of Assessments | 29 |
| Table 2 | NRX-101 Dose Titration | 32 |
| Table 3 | Lurasidone Dose Titration | 32 |
| Table 4 | NRX-101 Blinded Kits | 33 |
| Table 5 | Lurasidone Blinded Kits | 34 |
| Table 6 defined. | MADRS-10 Change From Baseline Outcomes: T-tests Error! Boo | kmark not |
| 4.2 List | t of Figures | |
| Figure 1 | DCS vs. Placebo for Treatment of Depression | 20 |

| Figure 2 | Randomization to NRX-101 vs. lurasidone following stabilization with ketamine . | 21 |
|---|---|---|
| Figure 3 | Study Schema | 23 |

### 5. ABBREVIATIONS

| Table of Abbreviations | Full Terms |
|---|---|
| ACPC | Aminocyclopropanecarboxylic Acid |
| AE | Adverse Event |
| SSIB | Subacute Suicidal Ideation or Behavior |
| BARS | Barnes Akathisia Rating Scale |
| BDRM | Biostatistics Data Review Meeting |
| BID | Twice Daily |
| BMI | Body Mass Index |
| BPI | Bipolarity Index |
| BPRS(+) | Brief Psychiatric Rating Scale(+) |
| CFB | Change from Baseline |
| CFR | Code of Federal Regulations |
| CGI-SS | Clinical Global Impressions of Severity for Suicidality |
| CHF | Congestive Heart Failure |
| CHRT-C | Concise Health Risk Tracking-Clinician |
| CHRT-SR | Concise Health Risk Tracking-Self Report |
| CLIA | Clinical Laboratory Improvement Amendments |
| Cmax | Maximum Concentration |
| CNS | Central Nervous System |
| СР | Conditional Power |
| CRO | Contract Research Organization |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DCS | D-cycloserine |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders Fifth Edition |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| eGFR | Estimated Glomerular Filtration Rate |
| ECT | Electroconvulsive Therapy |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HbA1c | Glycosylated Hemoglobin |
| HDPE | High Density Polyethylene |

| Table of Abbreviations | Full Terms |
|------------------------|-----------------------------------------------------|
| HIPAA | Health Insurance Portability and Accountability Act |
| НРМС | Hydroxymethylcellulose |
| ICH | International Conference on Harmonisation |
| ITT | Intent-to-Treat |
| IUD | Intrauterine Device |
| IWRS | Interactive Web Response System |
| Lurasidone | Lurasidone HCl |
| LOCF | Last Observation Carried Forward |
| MADRS | Montgomery Asberg Depression Rating Scale |
| MDD | Major Depressive Disorder |
| MMRM | Mixed Model Repeated Measures |
| NMDAR | N-methyl-D-aspartate Receptor |
| NOS | Not Otherwise Specified |
| OSFED | Other Specified Eating Disorder |
| PCP | Phencyclidine |
| PRISE | Patient Rated Inventory of Side Effects |
| QTcF | Fridericia's Correction Formula |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SIBAT | Suicide Ideation and Behavior Assessment Tool |
| SNRI | Serotonin and Norepinepherine Reuptake Inhibitors |
| SOP | Standard Operating Procedure |
| SSRI | Selective Serotonin Reuptake Inhibitor |
| TB | Tuberculosis |
| TeCA | Tetracyclic Antidepressant |
| TTF | Time to Treatment Failure |

#### 6. INTRODUCTION

#### 6.1 Suicidal Ideation and Behavior in Bipolar Disorder

Bipolar Disorder (formerly known as manic depressive disorder) is a well-established psychiatric diagnosis, with a prevalence of about 2.6% in the United States (approximately 8.5 million people) (Kessler et al., 2005). The risk of subacute suicidal ideation or behavior (SSIB) is uniquely high in patients during bipolar depressive episodes, compared to those with major depressive disorder (MDD), thought disorders, and personality disorders. Lifetime suicide behavior occurs in 25% to 56% of people with bipolar disorder (Nierenberg et al., 2001). About 40% of the nearly 50,000 annual deaths from suicide in the United States are associated with bipolar disorder (Mahli et al., 2015). The overall rate of death by suicide among patients with bipolar disorder is 164 per 100,000 person years, compared to about 14 per 100,000 person years for the general population. Those who have attempted suicide are 2.3 times more likely to die by suicide compared to those without a suicide attempt (Coryell et al., 2016). Thus, bipolar depression with suicidal ideation has uniquely lethal clinical characteristics (Pompili, et al., 2013).

#### **6.2** Current Treatment Options

Despite its lethal characteristics, there is no approved pharmacologic treatment for patients with bipolar depression and suicidal ideation. Electroconvulsive therapy (ECT), often combined with inpatient psychiatric care, remains the only Food and Drug Administration (FDA)-approved treatment for patients with acute suicidal ideation in bipolar depression, despite ECT's well-documented side effects that include memory loss and confusion, along with its high cost. However, the toxicity of ECT is such that it is less likely to be used in patients with subacute levels of suicidal ideation and no oral medication has been shown to reduce suicidal ideation in patients with depression in general or bipolar depression in specific. Physicians are increasingly cautious about the use of selective serotonin release inhibitors (SSRIs), particularly in patients with suicidal ideation because of evidence that SSRIs and other antidepressants may actually increase the risk of suicidal ideation, particularly in younger patients (Stone et al., 2009). This evidence has resulted in an FDA warning on the label of current antidepressants. Moreover, it seems clear that antidepressants do not decrease SSIB in proportion to their mitigating effect on symptoms of depression.

In recent years, several combined D2/5-HT2A antagonists have shown efficacy in treating bipolar depression (olanzapine/fluoxetine combination, quetiapine, and lurasidone) with treatment guidelines endorsing common use as first-line standard of care treatment in acute bipolar depression. While these medications are effective at reducing overall symptoms of depression, they do not specifically reduce suicidal ideation, as shown in recent clinical trials of lurasidone (Loebel et al., 2014a; Loebel et al., 2014b). Moreover, in these two studies, individuals with active suicidal ideation (Montgomery Asberg Depression Rating Scale [MADRS] item  $10 \ge 4$ ) were specifically excluded because of concerns regarding the possibility of exacerbating suicidality with

these medications. Similarly, acutely suicidal patients are routinely excluded from clinical trials of other experimental anti-depressive agents. Thus, bipolar depression with suicidal ideation represents a major unmet medical need that must frequently be treated with voluntary or involuntary hospitalization under highly supervised conditions and ECT.

#### 6.3 Preclinical Models of Anxiety and Akathisia

Although the mechanisms mediating antidepressant-related increases in suicide remain unclear, leading theories suggest that increases in anxiety/akathisia may play a critical role (Harada et al., 2014; Popovic et al., 2015). Serotonin-related anxiety/akathisia may be modeled in rodents using several well-established assay systems, such as the elevated plus maze, and are known to be sensitive to serotonergic agents (Sachdev and Brune, 2000). In this assay, reduced percent time spent in the open arms of the maze is believed to be associated with increased akathisia and anxiety. In contrast, increased total distance traveled in the maze is thought to be a signal related to psychosis. As shown by Javitt (2014), D-cycloserine (DCS) significantly reduces the anxiogenic effects of lurasidone and quetiapine, as measured by time spent in open arms, suggesting that this treatment might reduce medication-induced suicidality, as well as suicidality associated with bipolar depression itself.

Preclinical data, using the Rodent Akathisia model, suggests a potential synergistic interaction between DCS and lurasidone. On one hand, as described above, DCS appears to block the anxiogenic effects of lurasidone. On the other hand, lurasidone may reverse low-level psychotomimetic effects of DCS. Lurasidone mediates its antipsychotic effects at both D2 and 5-HT2A receptors. As opposed to pure serotonergic agents used in the treatment of major depressive disorders (e.g., SSRIs), the additional D2 blockade of lurasidone makes it a clinically effective antipsychotic; thus, it could also be effective in treating the psychotic symptoms that may be induced by an N-methyl-D-aspartate receptor (NMDAR) antagonist.

Clearly, the phenomena observed in rodents should not be viewed as isomorphic with drug-induced akathisia and/or restlessness/anxiety syndrome in humans. However, these findings provide a rationale for combining glycine site-binding NMDAR antagonists with 5-HT2A antagonists in phase 2 and 3 studies of otherwise-safe drugs for the treatment of bipolar depression. This is particularly true in situations where akathisia is believed to predispose vulnerable patients to suicide.

#### 6.4 Clinical Experience with DCS

Antidepressant effects of high-dose DCS were first noted in the late 1950s, when it was introduced as a treatment for tuberculosis (TB). Several clinicians noted dramatic improvement in patients' depressive symptoms, leading to suggestions of DCS' potential psychotropic effects. These effects were subsequently confirmed in small-scale clinical studies (Crane, 1959 and 1961). The mechanism of action was unknown at the time, and the finding was not pursued. The interaction of DCS with the NMDAR was first demonstrated in 1989 (Hood et al., 1989), leading to some

NRX-101 003  09 NOVEMBER 2023

interest in NMDAR blockers as potential antidepressant treatments (Trullas and Skolnick, 1990; Skolnick et al., 1996). For example, both DCS and the related compound aminocyclopropanecarboxylic acid (ACPC) were shown to be active in mice, using the forced swim test for depression (Lopes et al., 1997). To the best of our knowledge, no clinical antidepressant research programs targeting the NMDA receptor were initiated at that time.

Interest in the potential clinical use of DCS as an antidepressant agent was renewed following Berman's fortuitous observation of ketamine's rapid antidepressant effect (Berman et al., 2000). An initial study performed with DCS at a dose of 250 mg/day did not show therapeutic effects, but it did demonstrate a relative lack of psychotomimetic side effect when DCS was combined with concurrent antidepressant treatment (Heresco-Levy et al., 2006). Based upon these safety data, a study using a higher dose of 1000 mg/day was initiated, with results reported in 2013 (Heresco-Levy et al., 2013). At the higher dose of 1000 mg/day, significant beneficial effects were observed in 13 subjects vs. placebo control with SSRI-nonresponsive depressive symptoms. The improvements were manifested within 2 weeks and persisted throughout the 6-week treatment period. These data suggest a >0.9 effect size. In that study, a slow DCS titration was used, with 250 mg/day for 3 days, followed by 500 mg/day for 18 days (i.e., until the end of week 3); followed by 750 mg/day for 1 week (i.e., until the end of week 4), followed by 1000 mg/day (i.e., until the end of study). A statistically significant improvement was observed in the DCS group compared to placebo by the end of week 4, i.e., within 1 week of initiation of a DCS dose >500 mg/day (see Figure 1).

D-cycloserine (no Ketamine) delayed effect, sustained duration 30 Hamilton depression rating 25 20 scale (HDRS) 15 D-cycloserine (n=13) 10 Placebo (n=13) 5 2 6 0 4

Figure 1 DCS vs. Placebo for Treatment of Depression

Source: Heresco-Levy et al., 2013

The data above provided initial evidence that DCS may be useful as an NMDAR-targeted antidepressant, but the time of onset for DCS alone was suboptimal for treating acutely depressed individuals (Figure 1).

The data below provides evidence of efficacy from a study of NRX-101 versus Lurasidone in patients with severe bipolar depression (MADRS  $\geq$  30) and Acute Suicidal Ideation or behavior (C-SSRS 4, or 5), after an initial stabilization with a single infusion of ketamine.

Figure 2 Randomization to NRX-101 vs. lurasidone following stabilization with ketamine



Source: Javitt et. al. 2018

#### 6.5 Investigational Therapy

In accordance with FDA experience with lurasidone being used to successfully treat depression in bipolar disorder, participants will be randomized on Day 1 in a 1:1 ratio (NRX-101:lurasidone + placebo) and will receive maintenance treatment with matched twice-daily oral capsules. Participants will continue oral therapy through Day 42, according to treatment assignment.

It is anticipated that participants will also be receiving concurrent bipolar disorder—directed treatment with various predefined combinations of medications. This treatment regimen will be maintained upon entry into the study. However, any use of lurasidone, quetiapine, aripiprazole, risperidone, brexpiprazole, olanzapine, cariprazine, or lumateperone, will be discontinued at study entry. The treating psychiatrist should ensure that any medications to be discontinued can be done so safely. At entry, at the discretion of the investigators or the delegated treating physician subjects may continue their mood stabilizers which should not change over the course of the trial. In addition, participants receiving olanzapine/fluoxetine combination will continue to receive the fluoxetine component.

#### 6.6 Dose Selection

Lurasidone is an FDA-approved medication for depressive episodes associated with Bipolar I Disorder (bipolar depression) as monotherapy and as adjunctive therapy with lithium or valproate at doses of 20 mg to 120 mg daily. The target dose of 66 mg/day is based on the mean daily dose

of lurasidone observed during the fixed titration phase of the lurasidone registration trial for its indication in bipolar depression (Loebel et al., 2014b) and further validated in the STABIL-B trial (Javitt, et. al. 2018). Up-titrations are permitted if needed to doses of 99 or 132 mg/day, and down-titrations are permitted to 33 or 49.5 mg/day, which span the range of doses used in clinical studies of lurasidone (Loebel et al., 2014a; Loebel et al., 2014b).

DCS is well tolerated as a second-line treatment for TB at therapeutic split daily oral doses in the range of 500 to 1000 mg/day. Based on prior clinical results and animal studies, it is anticipated that therapeutic effects of DCS will be associated with plasma doses in excess of 25  $\mu$ g/mL, which in turn are generally associated with daily oral doses in excess of 10 mg/kg (i.e., 700 mg/day for a 70 kg) individual. A starting daily dose at 700 mg DCS and 33 mg lurasidone will be used, and then titrated over 2 days to the target dose of 950 mg DCS and 66 mg lurasidone. Down-titrations of DCS to 825 or 700 mg/day are available in the case of side effects to permit reduced dosing within the anticipated therapeutic range (700 – 950 mg/day). The maximum dose of 950 mg/day is within FDA-approved dosing limits for DCS.

#### 7. OBJECTIVES

#### 7.1 Primary Objective

The primary objective of the study is:

• To test the hypothesis that treatment with NRX-101 is superior to lurasidone (a standard of care medicine) in improving symptoms of depression as measured by the Montgomery Åsberg Depression Rating Scale (MADRS-10) total score in participants with severe bipolar depression and subacute suicidal ideation or behavior (SSIB).

#### 7.2 Key Secondary Objectives

- To test the hypothesis that NRX-101 is superior to lurasidone in reducing suicidal ideation or behavior as measured by the Clinical Global Impression of Severity of Suicidality Scale (CGI-SS)
- To test the hypothesis that NRX-101 is superior to lurasidone in time to treatment failure as defined as: study discontinuation due to adverse events; psychiatric hospitalization; or requiring a change in antidepressant treatment

#### 7.3 Additional Secondary Objectives

- To test the hypothesis that treatment with NRX-101 is superior to standard of care (lurasidone) in reducing suicidal ideation (MADRS item 10)
- To test the hypothesis that treatment with NRX-101 is superior to lurasidone in reducing the frequency of suicidal thoughts, suicidality and risk (SIBAT Module 7)
- To test the hypothesis that treatment with NRX-101 is superior to treatment with lurasidone in the subgroup of participants recently (i.e. within two weeks of enrollment)

treated with approved medications for bipolar depression (olanzapine/fluoxetine, quetiapine, cariprazine, lumateprone, or lurasidone).

#### 7.4 Safety Objectives

- To test the hypothesis that treatment with NRX-101 is superior to lurasidone (a standard of care drug) in reducing suicidality in depressed bipolar participants with SSIB, as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
- To test the hypothesis that participants treated with NRX-101 are less likely to suffer from akathisia than those treated with lurasidone as measured by the Barnes Akathisia Rating Scale (BARS)
- To test the hypothesis that fewer participants treated with NRX-101 will be discontinued for lack of efficacy or exacerbation of suicidality than participants treated with lurasidone.

#### 7.5 Overview

This is a group sequential, multicenter, randomized, double-blind, parallel-group, two-arm study comparing NRX-101 (n=37) to lurasidone (n=37) in a 1:1 ratio for the treatment of bipolar depression in participants with subacute levels of suicidal ideation, as reflected by the patient answering "yes" to item 3 and 4 on the C-SSRS within 4-weeks of screening, and do not require hospitalization.

Participants will be screened to ensure study eligibility prior to randomization on Day 1. Randomized participants will take either oral NRX-101 or lurasidone and placebo, in accordance with their treatment assignment, for 42 days. Participants will return to the investigational site on Day 70 for a follow-up visit (see Study Schema, Figure 3). During these visits, multiple psychometric scales will be completed, and participants will be assessed for safety, including the risk of increase in depression or suicidal ideation to the point where inpatient care or an alternative treatment is indicated.

Figure 3 Study Schema



#### 8. SELECTION OF PARTICIPANTS

Participants must meet all of the inclusion and none of the exclusion criteria to be qualified to participate in this study.

#### 8.1 Inclusion Criteria

- 1. 18 to 65 years of age, inclusive, at Screening.
- 2. Able to understand and provide written and dated informed consent prior to screening.
- 3. Deemed likely to comply with the study protocol, including communication of adverse events (AEs) and other clinically important information, including adherence to the text messaging component of the trial.
- 4. Will follow medical directions for psychiatric care, as appropriate, per the standard of care.
- 5. Resides in a stable living situation. A stable living situation will be defined as a minimum of 3 months at the same address with a reasonable expectation that the situation will continue such that the patient's ability to participate in the study will not be affected. Please note that housing in a shelter of any kind will not be deemed stable housing.
- 6. Previously diagnosed and treated for Bipolar Disorder (BD) I or II according to the criteria defined in the DSM-V.
- 7. Has an identified reliable informant/care partner, that is willing to provide information and/or supportive care as necessary.
- 8. The diagnosis of BD will have been made by a psychiatrist or other qualified licensed psychiatric provider able to render a diagnosis and be supported by the MINI 7.0.2.
- 9. Treatment with a medication indicated for use in bipolar disorder in the past five years (See Appendix 4 for list).
- 10. Confirmed active suicidal ideation (without the intention to act) as evidenced by an answer of 'Yes' on item 3 and/or 4 and not requiring hospitalization at Screening and an answer of 'No' on item 5 of the C-SSRS within 4-weeks of Screening.
- 11. A total score greater than or equal to 30 on the 10 items of the MADRS.
- 12. No co-morbidities, as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and electrocardiogram (ECG) which might interfere with compliance or the ability to assess efficacy or safety.
- 13. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following criteria, and agrees to continue use of the same method of birth control for the duration of study participation:

- a. Non-childbearing potential: physiologically incapable of becoming pregnant (i.e. permanently sterilized [status post-hysterectomy, bilateral tubal ligation] or post-menopausal with last menses at least one year prior to screening); or
- b. Childbearing potential, and meets the following criteria:
  - i. Use of any form of hormonal birth control for at least 2 months prior to Screening, on hormone replacement therapy that started prior to 12 months of amenorrhea, using an intrauterine device (IUD) for at least 1 month prior to Screening, in a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.
  - ii. Negative urine pregnancy test at Screening, confirmed by a second negative urinary pregnancy test at Day 1, prior to receiving any study treatment.
- 14. Body mass index (BMI) between 18-40 kg/m<sup>2</sup>; BMI up to 45 kg/m<sup>2</sup> is allowed with Medical Monitor review and approval.
- 15. If receiving concurrent psychotherapy, the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation.
- 16. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, maximum 2mg/daily, or trazodone) will be allowed if the therapy has been stable for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
- 17. Concurrent treatment with benzodiazepines is allowed up to a maximum dose 2mg/daily used for anxiety if therapy has been stable relative to dose and schedule for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study.
- 18. If women are receiving hormone replacement therapy or estrogen replacement, the therapy has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation.

#### 8.2 Exclusion Criteria

- 1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
- 2. Female who is pregnant or breastfeeding.
- 3. Female with a positive pregnancy test at Screening or prior to randomization.

- **4.** Current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to Screening. (Note: Substance use disorder cannot be the precipitant for study entry).
- **5.** A lifetime history of
  - a. phencyclidine (PCP)/ketamine drug abuse, or
  - b. failed use of ketamine for depression or suicidality.
- 6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
- 7. History of anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified (NOS), or other specified feeding and eating disorders (OSFED) within 3 years of Screening.
- 8. Has dementia, delirium, amnestic, or any other cognitive disorder.
- 9. Current major psychiatric disorder, diagnosed at Screening with the MINI 7.0.2 which is the primary focus of treatment, with bipolar disorder as the secondary focus of treatment, within the past 6 months.
- 10. Estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m<sup>2</sup> using the Cockcroft-Gault formula.
- 11. A clinically significant abnormality on the Screening physical examination that may affect safety or study participation, or that may confound interpretation of study results according to the study clinician.
- 12. Current episode of:
  - a. Myocardial infarction within 1 year of Screening.
  - b. Diagnosis of angina pectoris.
  - c. Prolonged QTc interval, as measured by Fridericia's correction formula (QTcF)
     ≥450 msec at Screening for males or ≥ 470 msec for females on 2 of 3
     measurements at least 15 minutes apart prior to randomization on Day 1.
- 13. Diagnosis of chronic lung disease, excluding asthma.
- 14. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS.
- 15. History of significant head trauma within the past two years.
- 16. Diabetes mellitus fulfilling any of the following criteria:

- Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 % at Screening.
- b. Admitted to the hospital for treatment of diabetes mellitus or diabetes mellitus—related illness in the past 12 weeks.
- c. Not under physician care for diabetes mellitus.
- d. Not on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to Screening.
- e. Not on the same dose of oral thiazolidinediones (glitazones) for the 8 weeks prior to Screening.
- 17. Any current or past history of any physical condition which, in the opinion of the investigator, may put the patient at risk or interfere with study results interpretation.
- 18. Diagnosis of HIV/AIDS.
- 19. Diagnosis of Hepatitis C.
- 20. On exclusionary concomitant psychotropic and non-psychotropic medications (see Appendix 1).
- 21. Prescribed more than one agent in each of the following categories at randomization:
  - a. Approved SSRIs.
  - b. Approved serotonin and norepinephrine reuptake inhibitors (SNRIs).
  - c. Approved tetracyclic antidepressants (TeCAs).

Note: Any/all 5hT2A medications will be discontinued at study entry. Participants currently on Lurasidone will be randomized to either standard of care or NRX\*-101 at the indicated starting dose.

- 22. Currently prescribed oxcarbazepine or carbamazepine.
- 23. Exclusionary laboratory values or any other clinically significant abnormal laboratory result (as determined by the investigator and Medical Monitor) at Screening.
- 24. Known allergies to lurasidone or Latuda<sup>®</sup>, cycloserine or Seromycin<sup>®</sup>, or the following excipients: mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or hydroxypropylmethylcellulose (HPMC).
- 25. Participation in any clinical trial with an investigational drug or device within the past month or planned concurrent study participation.
- 26. Study site personnel and/or persons employed by NRx Pharma, Inc., the Contract Research Organization (CRO), the investigator, or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate

- family member (i.e., spouse, parent, child, or sibling [biological or legally adopted]) of such persons.
- 27. Positive urine toxicity screening for use of any cocaine, opiates and non-prescribed amphetamine and non-prescribed barbiturates (Note: Cannabinoids or Marijuana use is not exclusionary unless the patient meets the criteria for cannabis withdrawal).
- 28. Signs and symptoms of active or residual COVID-19, or unresolved symptoms of COVID-19 that impact health, e.g. requirements for oxygen supplementation, etc. Discharge from an inpatient hospitalization for more than 48 hours for COVID-19 within the past 28 days.

#### 9. STUDY VISITS

#### 9.1 Study Visits

Study subjects are required to undergo the below frequency of assessments, 2 of which can be done by video / conference if required due to COVID-19 circumstances. Investigators may always conduct unscheduled visits to monitor subject safety. The schedule of assessments is synchronous with the main protocol and congruent with monitoring participants of lesser acuity.

A schedule of study visits and assessments is provided in Table 1.

 Table 1
 Schedule of Assessments

| | Screening Treatment | | | | | | Follow up <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Study Day | Day<br>-10 to -1 | Day 1 <sup>2</sup><br>Baseline | Day 7 | Day 14 <sup>3</sup> | Day 28 <sup>3</sup> | ET/Day 42 <sup>3</sup> | Day 70 |
| Informed Consent | X | | | | | | |
| Eligibility Review | X | X | | | | | |
| Randomization | | X | | | | | |
| Demographics | X | | | | | | |
| Medical History | X | | | | | | |
| Psychiatric History | X | | | | | | |
| MINI | X | | | | | | |
| MINI Severity/Disability | | X | | | | X | |
| Subject Eligibility | X | X | | | | | |
| Physical Exam <sup>4</sup> | X | | | | | X | |
| Vital Signs, Weight <sup>5</sup> | X | X | | X | X | X | |
| ECG <sup>6</sup> | X | X | | | | X | |
| Pregnancy Test (Urine dipstick) | X | X | | | | | |
| Drugs of Abuse Screen (Urine dipstick) <sup>7</sup> | X | X | X | X | X | X | |
| Fasting Chemistry,<br>Hematology | X | | | | | X | |
| C-SSRS <sup>8</sup> | X | X | X | X | X | X | |
| MADRS | X | X | X | X | X | X | |
| CGI-SS | X | X | X | X | X | X | |
| CHRT-C, -SR | X | | X | X | X | X | |
| BPRS psychosis subscale | X | X | X | X | X | X | |
| BARS 12 | X | X | X | X | X | X | |
| PRISE | X | X | X | X | X | X | |
| Adverse Events | | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X |
| Adherence device training <sup>9</sup> | | X | | | | | |
| Dispense investigational product and review adherence <sup>10</sup> | | Х | X | X | X | | |
| Site monitoring of adherance <sup>11</sup> | | | X | X | X | X | |

Follow up visit will be a phone call; the study visit may occur within ± 7 days of the scheduled day (anchored to the Day 1 visit).

<sup>&</sup>lt;sup>2</sup> Day 1 procedures need to meet eligibility criteria and will be performed prior to first dose.

<sup>&</sup>lt;sup>3</sup> Study visits occurring after Day 7 may occur within ± 3 days of the scheduled day (anchored to the Day 1 visit). Study visits 3, 4, 5, 7 may be done virtually, preference is through videoconference.

<sup>&</sup>lt;sup>4</sup> Full physical exam (including a neurological exam and height) at Screening and Visit 6 will be performed, and a brief exam (Blood Pressure, Respiration Rate, Heart Rate, and Temperature) will be performed at subsequent time points.

<sup>&</sup>lt;sup>5</sup> After 5 min at rest, supine or sitting systolic and diastolic blood pressure and heart rate are recorded at each indicated visit. Weight is measured only at Screening and Visits 2,4,5, and 6.

<sup>&</sup>lt;sup>6</sup> 12-lead ECG.

Subjects who have 2 consecutive positive urine screens should be withdrawn from study, in case of a subject not being able to visit a site due to COVID-19 restrictions or impediments arrangements should be made for an outpatient test, or the investigators should note this and make an assessment during the tele visit, annotation should be included in the EDC why the drug screen text could not be done. In the case where the subject has 2 consecutive negative urine screens, the subject can skip

- the next urine screen. Investigators can bring the subject in for a urine screen at any time if suspected drug use. Note: Since Cannabis use is not exclusionary, a positive UDS will not require that patient be withdrawn from the study.
- 8 "Baseline" version should be administered at screening and "Since Last Visit" version should be administered at all other time points.
- Adherence device training should be performed pre-dose on Day 1 or with the first dose. Additional training will be provided as necessary. The subject's cellphone number will be input in a secure field of the EDC by the study site personnel, this field will only be accessible to designated study site personnel. The system will send a text message at designated hours to the subject as a reminder to take study the medication. The subject must respond affirmatively to enable compliance tracking. Absence of a response or a negative response will trigger a notification to the site.
- <sup>10</sup> Medication adherence will be reviewed and returned pills recorded.
- 11 Sites will monitor / review compliance for a target goal of 85 percent compliance of all doses taken. If more than 2 consecutive doses are missed they should contact the subject and counsel the subject on the need for compliance before the next scheduled dose.
- <sup>12</sup> Rating akathisia using BARS needs to be a video call if completed remotely and will be documented.

#### 9.1.1 Screening Period

Once a patient agrees to participate in the study, indicated by signing the informed consent form, the patient is admitted to the study. A full medical and psychiatric history will be taken, and a physical and laboratory examination will be performed, as outlined in the Schedule of Assessments (Table 1). The Screening period may extend to 10 days following the signing of the informed consent form in order to allow sufficient time for Screening procedures to be completed and results reported.

#### 9.1.1.1 Rating Scale

The site will upload digital audio files and score summaries of the MINI and MADRS, and the score summary for the C-SSRS. The MINI diagnostic interview, MADRS, and C-SSRS scores will be reviewed by an Expert Psychometrician for all study participants.

#### 9.1.1.2 eGFR Calculation

Using the results of the chemistry panel, glomerular filtration rate will be estimated by using the creatinine clearance value calculated using the Cockgroft-Gault formula, as follows:

- CrCl (male) = ( $[140\text{-age}] \times \text{weight in kg}$ )/(serum creatinine  $\times 72$ )
- CrCl (female) = CrCl (male)  $\times$  0.85

Because participants with renal insufficiency may accumulate cycloserine, participants with moderate renal insufficiency (eGFR < 60 ml/min/1.73 m<sup>2</sup>) or worse will be excluded from study participation.

#### 9.1.1.3 Screen Failures

In the event a patient is a screen failure, the patient may be rescreened at the discretion of the investigator and Medical Monitor.

#### 9.1.2 Treatment and Follow-up Periods

Participants that continue to meet MADRS and C-SSRS eligibility will be randomized to receive the first dose of blinded treatment on Day 1. This visit will be followed by Treatment Period visits at Days 7, 14, 28, and 42. Following completion of the Treatment Period, participants will be

contacted via telephone for follow-up on Day 70. In order to allow scheduling flexibility, and (considering pandemic related limitations), visit windows will be allowed as noted in Table 1. Participants will be withdrawn from the study if their urine toxicology screenings at two consecutive study treatment visits are positive for cocaine, opiates, non-prescribed amphetamines, or non-prescribed barbiturates.

#### 9.1.3 Early Termination Visit

Every effort will be made to keep the participants in the study for the full study period. However, if a patient decides to discontinue the investigational product, the patient will be asked about the reason(s) for discontinuation and the presence of any AEs. If possible, the patient will be asked to complete the Day 42/Early Termination (ET) visit prior to discontinuation, and day 70 to assess safety. Following completion of the Early Termination Visit, the patient will either be treated by the investigator with standard of care or, should the patient choose, return to treatment by a prior/referring physician. In this case, the investigator will facilitate and coordinate follow-up to ensure continuity of care.

Participants who discontinue from the study will not be replaced.

#### 10. TREATMENT OF PARTICIPANTS

#### 10.1 Investigational Drug Dose and Administration

Participants will be instructed to take all oral investigational product with food. Participants will be trained to ingest food prior to or immediately after ingestion of investigational product, and they will be reminded of this requirement at each study visit as part of adherence monitoring.

Participants should be instructed to avoid eating grapefruit or drinking grapefruit juice while on study as it may affect the amount of medication in the blood. This fruit and its juice can raise blood levels of some antipsychotic drugs such as lurasidone.

#### **10.2 Investigational Product**

NRX-101 is a capsule intended for oral administration. Each NRX-101 capsule contains DCS and lurasidone HCl. Inactive ingredients include mannitol, croscarmellose sodium, silica dioxide, and magnesium stearate.

The physical description and composition of each capsule is described in the Investigator Brochure. NRX-101, lurasidone, and placebo capsules are matched in terms of size, shape, and color with no discernible difference in appearance or physical description. The lurasidone capsules contain lurasidone at the same dosage as the matched NRX-101 capsules.

#### 10.3 Investigational Product Titration

Investigators will have the ability to increase the lurasidone dose at any point after the initial titration period for control of agitation or psychotic symptoms, or to decrease both the DCS and lurasidone dose in response to somnolence. No other dose modifications will be allowed.

Titrations of investigational product will be affected while maintaining a blinded study design (see Table 2 for NRX-101 and Table 3 for lurasidone). Up-titration will increase the lurasidone dose, and will not alter the DCS dose. Down-titration decreases the total daily dose of both lurasidone and DCS in the NRX-101 group and only the lurasidone dose in the lurasidone group.

**Table 2** NRX-101 Dose Titration

| | Morning Dose (mg) | | Evening Dose (mg) | | Total Daily Dose (mg) | |
|---|---|---|---|---|---|---|
| Day | DCS | Lurasidone | DCS | Lurasidone | DCS | Lurasidone |
| 1 | 350 | 16.5 | 350 | 16.5 | 700 | 33 |
| 2 | 475 | 33 | 475 | 33 | 950 | 66 |
| 3 | 475 | 33 | 475 | 33 | 950 | 66 |
| 4 | 475 | 33 | 475 | 33 | 950 | 66 |
| 5 | 475 | 33 | 475 | 33 | 950 | 66 |
| Maintenance Dose | 475 | 33 | 475 | 33 | 950 | 66 |
| Up-titration (if needed) | | | | | | |
| step 1 | 475 | 33 | 475 | 66 | 950 | 99 |
| step 2 | 475 | 66 | 475 | 66 | 950 | 132 |
| Down-titration (if needed) | | | | | | |
| step 1 | 350 | 16.5 | 475 | 33 | 825 | 49.5 |
| step 2 | 350 | 16.5 | 350 | 16.5 | 700 | 33 |

**Table 3** Lurasidone Dose Titration

| | Morning | Morning Dose (mg) | | Evening Dose (mg) | | y Dose (mg) |
|---|---|---|---|---|---|---|
| Day | DCS | Lurasidone | DCS | Lurasidone | DCS | Lurasidone |
| 1 | 0 (placebo) | 16.5 | 0 (placebo) | 16.5 | 0 (placebo) | 33 |
| 2 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| 3 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| 4 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| 5 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| Maintenance Dose | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| Up-titration (if needed) | | | | | | |
| step 1 | 0 (placebo) | 33 | 0 (placebo) | 66 | 0 (placebo) | 99 |
| step 2 | 0 (placebo) | 66 | 0 (placebo) | 66 | 0 (placebo) | 132 |
| Down-titration (if needed) | | | | | | |
| step 1 | 0 (placebo) | 16.5 | 0 (placebo) | 33 | 0 (placebo) | 49.5 |
| step 2 | 0 (placebo) | 16.5 | 0 (placebo) | 16.5 | 0 (placebo) | 33 |

# 11. INVESTIGATIONAL PRODUCT MATERIALS AND MANAGEMENT

#### 11.1 Packaging and Labeling

Investigational product will be supplied in high-density polyethylene (HDPE) bottles with a foil induction seal and screw-top closures. Each bottle will contain two capsules, the required dose for either morning or evening administration, as well as a desiccant to aid stability. The bottles will be packaged into a cardboard kit containing two bottles for each day.

Six kit types will be available for each patient. Kit 1 will contain a 7-day titration pack consisting of 14 bottles, each containing two capsules, for use during the first 7 days of the study (+2 days). Kits 2 to 5 will contain three-day step-up or step-down packs with six bottles, each containing two capsules and will only be dispensed if the patient requires a dose titration. Kit 6 will contain a 7-day maintenance dose pack with 14 bottles, each containing two capsules. A description of the six kit types are provided in Table 4 for NRX-101 and in Table 5 for lurasidone.

Table 4 NRX-101 Blinded Kits

| Kit Type | Day | Morning Dose (mg) | | Evening Dose (mg) | | Total Daily Dose (mg) | |
|---|---|---|---|---|---|---|---|
| | | DCS | Lurasidone | DCS | Lurasidone | DCS | Lurasidone |
| 1 (7 Days) | 1 | 350 | 16.5 | 350 | 16.5 | 700 | 33 |
| | 2 | 475 | 33 | 475 | 33 | 950 | 66 |
| | 3 | 475 | 33 | 475 | 33 | 950 | 66 |
| | 4 | 475 | 33 | 475 | 33 | 950 | 66 |
| | 5 | 475 | 33 | 475 | 33 | 950 | 66 |
| | 6 | 475 | 33 | 475 | 33 | 950 | 66 |
| | 7 | 475 | 33 | 475 | 33 | 950 | 66 |
| | Up- | | | | | | |
| | titration | | | | | | |
| 2 (3 Days) | step 1 | 475 | 33 | 475 | 66 | 950 | 99 |
| 3 (3 Days) | step 2 | 475 | 66 | 475 | 66 | 950 | 132 |
| | <b>Down-titration</b> | | | | | | |
| 4 (3 Days) | step 1 | 350 | 16.5 | 475 | 33 | 825 | 49.5 |
| 5 (3 Days) | step 2 | 350 | 16.5 | 350 | 16.5 | 700 | 33 |
| 6 (7 Days) | Maintenance | 475 | 33 | 475 | 33 | 950 | 66 |

NRX-101 003  09 NOVEMBER 2023

**Table 5** Lurasidone Blinded Kits

| Kit Type | Day | Morning Dose (mg) | | Evening Dose (mg) | | Total Daily Dose (mg) | |
|---|---|---|---|---|---|---|---|
| | | DCS | Lurasidone | | Lurasidone | DCS | Lurasidone |
| 1 (7 Days) | 1 | 0 (placebo) | 16.5 | 0 (placebo) | 16.5 | 0 (placebo) | 33 |
| | 2 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | 3 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | 4 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | 5 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | 6 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | 7 | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |
| | Up- | | | | | | |
| 2 (3 Days) | step 1 | 0 (placebo) | 33 | 0 (placebo) | 66 | 0 (placebo) | 99 |
| 3 (3 Days) | step 2 | 0 (placebo) | 66 | 0 (placebo) | 66 | 0 (placebo) | 132 |
| | Down-titration | | | | | | |
| 4 (3 Days) | step 1 | 0 (placebo) | 16.5 | 0 (placebo) | 33 | 0 (placebo) | 49.5 |
| 5 (3 Days) | step 2 | 0 (placebo) | 16.5 | 0 (placebo) | 16.5 | 0 (placebo) | 33 |
| 6 (7 Days) | Maintenance | 0 (placebo) | 33 | 0 (placebo) | 33 | 0 (placebo) | 66 |

Each investigational product label will include the following information:

- Name of sponsor and address
- Protocol number
- Number of capsules
- Storage conditions
- Investigational drug statement (for clinical trial use only)
- Drug packager lot number
- Kit/Medication number
- Contents
- Administration statement
- Bar code
- Child warning
- Grapefruit warning
- Spaces to record:
  - o Subject number
  - o Date dispensed

#### **11.1.1 Storage**

Investigational product will be stored at room temperature of 20°C to 25°C (68°F to 77°F); excursions will be permitted to 15°C to 30°C (59°to 86°F).

#### 11.1.2 Accountability

The clinical site is required to maintain current drug dispensation and accountability logs throughout the study. All unused supplies will be checked against the drug dispensation and accountability logs during the study and/or at the end of the study.

#### 11.1.3 Handling and Disposal

There are no special handling requirements for the investigational product. Unused investigational product will be returned to the drug depot for disposal.

Please refer to the Pharmacy Manual for further information.

#### 11.2 Study Drug Monitoring

An Electronic Patient Reported Outcome (ePRO) System will be used in this study. The ePRO will send daily reminders at designated hours to participants enrolled in the study to take their study drug via text messages to each patient's own cell phone. The patient must respond affirmatively to enable compliance tracking.

The ePRO system will also host an audit trail for recording patient responses and an email alert message system to the site staff if no response or negative response is received from the patient. The ePRO system will be available to authorized site users through the Prevail Single Interface <sup>TM</sup> (SI).

Patient will grant the study site permission to contact him/her on the mobile device if a personal telephone number(s) cannot be reached. Additionally, sites will review drug utilization through receipt of used drug kits and assessments with participants.

#### 12. EFFICACY ASSESSMENTS

Study procedures are described below. Assessment time points are included in the Schedule of Assessments (Table 1).

#### 12.1 Montgomery Asberg Depression Rating Scale (MADRS)

The Montgomery Åsberg Depression Rating Scale is a 10-item clinician-rated scale, with each item rated on a 0–6 severity scale (Montgomery, Åsberg 1979). The timeframe for the baseline MADRS-10 recorded at Screening and Day 1 is the past seven days; for the MADRS-10 recorded at all time points thereafter, the timeline measured will be since the last assessment.

#### 12.2 Clinical Global Impression-Severity for Suicide

The three Clinical Global Impression scales represent the final three global ratings from the Suicidality Ideation Inventory and Behavior Assessment Tool (SIBAT Module 7), which is designed for the clinician to assess the relative risk and overall risk of suicide across different time scales (Alphs et al., 2016). The questions assess the clinician's global impression of immediate risk of suicide (that day), imminent risk of suicide (over the next 7 days), and long-term risk (i.e., likely to end their life by suicide sometime in the future). Each risk (immediate, imminent, long-term) is rated along a graded impressions scale starting at 0 ('normal', 'not suicidal' or 'no risk') and ranges to 6 ('among the most extremely suicidal' or 'extreme risk for imminent'/'long-term suicide').

#### 12.3 Brief Psychiatric Rating Scale (BPRS psychosis subscale)

Overall the Brief Psychiatric Rating Scale (BPRS) is an 18-item clinician-rated scale that assesses a range of psychotic and affective symptoms, rated from both observation of the patient and the patient's own report (Overall and Gorham, 1962). Only the 4-item positive symptom subscale referred to in this document as the "BPRS psychosis subscale" (i.e., suspiciousness, hallucinations, unusual thought content, and conceptual disorganization) will be used.

# 12.4 Concise Health Risk Tracking – Self Report (CHRT-SR) and Clinician Rating (CHRT-C)

The Concise Health Risk Tracking – Self Report (CHRT-SR) and – Clinician (CHRT-C) are assessments of suicidality and related thoughts and behaviors (Trivedi et al., 2011). The CHRT-SR is a 16-item self-report suicidal ideation scale, and the CHRT-C is a 9-item clinician-rated behavioral module. Items are rated on a fully anchored five-point Likert scale with responses ranging from 1 (strongly disagree) to 5 (strongly agree). The time frame is the past seven days.

#### 13. OTHER DIAGNOSTIC INSTRUMENTS

#### 13.1 Mini International Neuropsychiatric Interview (MINI) 7.0.2

The MINI (Sheehan et al., 1998) is a short, structured diagnostic interview developed initially in 1990 by psychiatrists and clinicians in the United States and Europe for DSM-III-R and ICD-10 psychiatric disorders. The tool has been updated to map to DSM-5 diagnostic criteria in the MINI 7.0.2.

#### 13.2 Bipolarity Index (BPI)

For this study, the BPI is integrated with the patient eligibility evaluation. The BPI (Aiken et al., 2015) is a clinician-rated scale that rates cardinal features of bipolar disorder across five domains: episode characteristics (signs and symptoms); age of onset (first episode); course of illness; response to treatment; and family history. Possible scores range from 0–100 and a score of 50 has
a high sensitivity and specificity for the identification of bipolar disorder. The index scores will not be used for study entry, but will help inform diagnostic impression.

## 14. ASSESSMENT OF EFFICACY

#### 14.1 Primary Efficacy Endpoint

The primary efficacy endpoint is:

• Mean change from baseline in total MADRS score

#### 14.2 Key Secondary Efficacy Endpoints

The key secondary efficacy endpoint are:

- Change from baseline over 42 days in CGI-SS
- Time to treatment failure in each arm

## 14.3 Additional secondary efficacy endpoints:

- Mean change from baseline in Suicidal Thoughts on the MADRS (MADRS item 10)
- Change from baseline to Day 14 in MADRS total score
- Change from baseline in each item of the Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 (clinical global impressions of frequency of suicidal thinking, severity of suicidality, and imminent and long-term risks)
- Change from baseline to endpoint (Day 42/exit) in MADRS total score in the subgroup of participants who were recently (within 2-weeks) on approved medications for bipolar depression
- Percent in remission at Day 42/exit.

## 15. ASSESSMENT OF SAFETY

Study procedures are described below. Assessment time points are included in the Schedule of Assessments (Table 1).

#### 15.1 Safety Scales

## 15.1.1 Columbia Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed in the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment (Posner et al., 2007). The timeframe for assessment is for both lifetime and the past 4-weeks for the Screening scale and since the last visit for all other ratings.

# 15.1.2 Patient Rated Inventory of Side Effects (PRISE)

The Patient Rated Inventory of Side Effects (PRISE) is a self-rated questionnaire (Rush and Asberg, 1999; Wisniewski et al., 2006) will be used to assess the specific symptoms considered by participants to be more or less tolerable drug side effects. The timeframe for assessment is at Screening for the Screening scale and in the past week for all other ratings.

# 15.1.3 Barnes Akathisia Scale (BARS)

The Barnes Akathisia (BARS) (Barnes, 1989) is a clinician-rated scale to assess drug-induced akathisia as absent, mild, moderate, or severe. It comprises items for rating the observable, restless movements which characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia. In addition, there is an item for rating global severity. The timeframe for the scale is "at this time."

#### 15.2 Adverse Events and Serious Adverse Events

#### 15.2.1 Definition of Adverse Events

An AE is any untoward medical occurrence in a clinical study patient administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship to the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.

This definition includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.

The following variables will be collected for each AE:

- AE (verbatim)
- The date and time when the AE started and stopped
- Maximum intensity or changes in intensity
- Whether the AE is serious or not (see Section 15.2.3)
- Expectedness
- Investigator assessment of relationship to investigational product
- Action taken with regard to the investigational product (uptitration, downtitration, temporarily discontinued, permanently discontinued or no action taken)

- AE caused patient's withdrawal from the study (yes or no)
- Outcome

Adverse events will be collected from the time of signature on the informed consent form throughout the Follow-up visit or early termination. Whenever possible, diagnoses will be given when signs and symptoms are due to a common etiology (e.g., cough, runny nose, sneezing, sore throat, and head congestion will be reported as "upper respiratory infection").

Worsening symptoms of the primary study condition (i.e., bipolar depression) will be recorded as a primary endpoint rating.

Any AE(s) that are unresolved at the follow-up visit (Day 70) will continue to be followed by the investigator for as long as medically indicated, but without further recording in the eCRF. The Contract Research Organization (CRO) and its representative retain the right to request additional information for any patient with ongoing AE(s)/SAE(s) at the end of the study, if deemed medically necessary.

#### 15.2.2 Adverse Event Intensity and Relationship

Intensities for each AE will be assessed by the investigator as:

- Mild: Awareness of sign or symptom, but easily tolerated;
- Moderate: Discomfort sufficient to cause interference with normal activities; or
- Severe: Incapacitating, with inability to perform normal activities.

Relationship to investigational product will be assessed by the investigator according to the following categories:

- Not Related: Clearly and incontrovertibly due only to extraneous causes and does not meet criteria listed under possible or probable.
- Unlikely Related: Does not follow a reasonable temporal sequence from administration.
   May have been produced by the patient's clinical state or by environmental factors or other therapies administered.
- Possibly Related: Follows a reasonable temporal sequence from administration but may have been also produced by the patient's clinical state, environmental factors, or other therapies administered.
- Related: Clear-cut temporal association with administration with improvement on cessation of investigational product or reduction in dose. Reappears upon re-challenge. Follows a known pattern of response to the investigational product.

#### 15.2.3 Recording of Adverse Events

AE(s) spontaneously reported by the patient in response to an open-ended question from study personnel, such as, "Have you had any health problems since the previous visit?" or that are revealed by observation will be recorded at each visit. When reporting AE(s), the recording of diagnosis is preferred (when possible), rather than reporting the list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be recorded separately.

Participants should be encouraged to contact the investigator or a member of the clinical site staff at any time between visits concerning AE(s)or worsening of symptoms.

#### 15.2.4 Definition of Serious Adverse Events

The following criteria define an SAE:

- Death
- Life-threatening event
- Inpatient hospitalization >24 hours or prolongation >24 hours of inpatient hospitalization
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect
- Medically important event, as defined in this protocol\*

\*Medical and scientific judgment will be exercised in deciding whether expedited reporting is also appropriate in other situations, such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above. These will usually be considered serious.

In addition, the following variables will be collected, where applicable, for SAEs:

- Date AE met criteria for SAE
- Date investigator became aware of SAE
- Description of SAE
- Explanation of seriousness of the AE
- Date of hospitalization
- Date of discharge
- Probable cause of death
- Date of death
- Autopsy performed

- Causality assessment in relation to investigational product
- Causality assessment in relation to other medication

It is important to distinguish between serious and severe AE(s). Severity is a measure of intensity, whereas seriousness is defined by these criteria. An AE of severe intensity need not necessarily be considered serious. If inpatient hospitalization results from worsening psychiatric symptoms or suicidal ideation, the hospitalization will be reported as an SAE.

SAEs will be reported from the time of informed consent through the Follow-up visit or early termination. Unsolicited SAEs will be collected up to 30 days after the last study treatment.

#### 15.2.5 Reporting Serious Adverse Events

When an SAE is discovered, it will be reported immediately (within 24 business hours of the site's knowledge of the event) to the Sponsor/CRO Medical Monitor. Reportable events which do not meet the criteria for an SAE will include (but will not be limited to): (a) pregnancy, and (b) clinically significant (in the judgment of the investigator) severe psychiatric complications.

The eCRF will provide a mechanism for sites to report SAEs, and for investigators and the Medical Monitor to sign off on the SAE reports.

Reportable SAEs will be sent to the FDA by the sponsor and sites will be notified. Sites are responsible for submission of SAE reports to their IRB(s), in accordance with IRB policies.

# 15.2.6 Anticipated Serious Adverse Events

Tan et al (2021) publication Identifying Anticipated Events of Future Clinical Trials by Leveraging Data from the Placebo Arms of Completed Trials looked at 18 Randomized, double-blind, controlled trials of Bipolar Depression that met similar inclusion and exclusion criteria to identify the most common Serious Adverse Events.

Based on this publication, the anticipated Serious Adverse Events are:

- Hospitalization, psychiatric symptoms
- Suicidal behavior, overdose
- Cholecystitis
- Fall
- Road traffic accident, injury

#### 15.2.6.1 Overdose

Overdose of the investigational product will be considered an SAE, even when there are no symptoms or additional AEs, and will be reported according to the guidelines in Section 15.2.5. An overdose associated with symptoms must be reported as an AE.

# 15.2.6.2 Suicidal Ideation and Clinical Management

The documentation and proper management of suicidal ideation by sites will be documented with the use of the C-SSRS, completed by site clinicians during all visits. Safety will be evaluated throughout the course of the study.

Any patient who, based on the investigator's judgment, poses an imminent risk of suicide should be discontinued from the study. Suicide risk is assessed by the clinician at every visit.

Suicide, self-harm, and attempted suicide, irrespective of the method, will be reported as AEs (all suicides are SAEs; attempted suicides are considered to be SAEs). The event will be identified as suicide or attempted suicide, and the method of the suicide or attempt will be provided. If an attempted suicide meets the criteria for an SAE, the event must be reported according to the guidelines in Sections 15.2.4. If a suicide attempt does not meet the criteria for an SAE, it will be considered a reportable AE, and a Suicidal Ideation or behavior Reportable Event Form will be completed by the investigator and submitted in accordance with the SAE reporting procedure in Section 15.2.5.

# **15.2.6.3 Pregnancy**

If a patient (or patient's partner) becomes pregnant during the study, it must be reported within 24 business hours of the time the investigator becomes aware of the event and in accordance with the procedures described on the Pregnancy Report Form. Although pregnancy itself is not regarded as an SAE/AE, unless there is a suspicion that a study drug may have interfered with the effectiveness of a contraceptive medication, the pregnancy details will be captured in the AE/SAE module of the eCRF. Any pregnancy that occurs from Visit 1 to 30 days following the last dose given will be followed for gestational outcome, and the outcome will be reported to the sponsor. The female patient will be discontinued from investigational product, but will continue to attend study visits for the duration of her participation in the study.

#### 15.3 Concomitant Medications, Therapies, and Alcohol Restrictions

#### 15.3.1 Concomitant Medications

Lurasidone is contraindicated with the use of strong CYP3A4 inhibitors (e.g., ketoconazole) and strong CYP3A4 inducers (e.g., rifampin) (see Appendix 1). The lurasidone dose should not exceed 40 mg/day if co-administered with moderate CYP3A4 inhibitors. There are no known reported interactions between DCS and lurasidone.

It is anticipated that participants entering the study will be receiving concurrent disorder-directed treatment with various combinations of medications, including:

 Approved antidepressants (e.g., SSRIs, SNRIs, TeCAs, fluoxetine), but not 5-HT-2A antagonists (lurasidone, aripiprazole, olanzapine/fluoxetine, quetiapine, cariprazine, or lumateperone) • Mood stabilizers (e.g., lithium, valproic acid, and lamotrigine)

Participants will be permitted into the study if they are treated with no more than one drug from each category of the indicated classes. Approved antidepressants and mood stabilizers will be maintained at stable dosages throughout the study. This is both to ensure continued treatment and to prevent withdrawal symptoms that may occur if such drugs are rapidly discontinued. Participants—taking aripiprazole, risperidone, brexpiprazole, lumateperone, olanzapine, cariprazine, or quetiapine will discontinue these medications prior to Randomization in order to avoid overlap with lurasidone.

Allowed concomitant medications include any prescription or over-the-counter medication not specifically excluded by the protocol (see Appendix 1), as well as stable, ongoing antidepressant or mood stabilizer therapy and stable allowed hypnotic therapy. Participants requiring excluded medications will be discontinued from the study and an Early Termination Visit will be performed in accordance with Section 9.1.3.

Prohibited concomitant medications that the patient and the investigator agree to discontinue for the purpose of study entry will be washed out for a period defined by the Investigator in consultation with the Medical Monitor. In the event concomitant medication washout is appropriate for a patient per investigator judgment, the patient must sign the informed consent form prior to beginning the washout period. Clinically appropriate tapering regimens should be used, if applicable. The Screening period may be extended, upon consultation with the Medical Monitor, to allow for a sufficient washout period.

All concomitant medications taken during the study and 4-weeks prior to study entry will be recorded in the electronic case report form (eCRF) for each patient, along with dosage information and start and stop dates.

#### 15.3.2 Concomitant Therapy

Participants receiving concurrent psychotherapy that has been stable in type and frequency (e.g., weekly, monthly) for at least 3 months prior to Screening are eligible for study entry if the psychotherapy is expected to remain stable for the duration of the patient's participation in the study. Any changes in psychotherapy type and/or frequency during the study should be discussed with the Medical Monitor as soon as the investigator is aware of the proposed change.

#### 15.3.3 Alcohol Restrictions

Participants should not use alcohol during the study. Ethyl alcohol may increase the possibility and risks of seizures in participants with a history of alcoholism receiving cycloserine.

#### 15.3.4 Positive Drug Screen

Participants who have a positive urine drug screen two times in a row for use of any cocaine, opiates and non-prescribed amphetamine and non-prescribed barbiturates will be withdrawn from the study.

# 15.4 Laboratory/Diagnostic Procedures

Clinical laboratory safety testing will be performed locally at the study site using a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. The frequency and type of procedures are detailed in the Schedule of Assessments (Table 1). Local laboratory normal ranges must be reported according to gender.

Participants will have their blood drawn for clinical chemistry (ALT, AST, GGT, ALK phosphatase, Creatinine, T4, T3,TSH, Albumin, BUN, Calcium, Sodium, Potassium, Chloride, Glucose, Total Bilirubin, Direct Billirubin, Total Protein, Total Cholesterol, HDL/LDL, Triglycerides, Uric Acid, HbA1c) and hematology testing (Red blood cell count, White blood cell count, Platelet count, Hemoglobin, Hematocrit, Neutrophils Absolute or percent, Lymphocytes Absolute or percent, Monocytes Absolute or percent, Eosinophils Absolute or percent, Basophils Absolute or percent). Urine sample testing for pregnancy and drug screen will be by dipstick. In the event of clinically significant abnormal laboratory test result(s), follow-up laboratory testing may be conducted, at the discretion of the investigator. If applicable, clinically significant changes from baseline in laboratory results will be noted as AE(s), in accordance with Section 15.2.1.

#### 15.5 Physical Examinations, Vital Signs, Height, and Weight

Physical examinations, vital signs, height, and weight will be obtained at the noted visits. Vital signs (blood pressure and heart rate) may be repeated 15 min apart, as needed, in order to obtain a resting reading. If applicable, clinically significant changes from baseline in physical examination parameters, vital signs, and weight will be noted as AE(s), in accordance with Section 15.2.1.

#### 15.6 Electrocardiograms

Twelve-lead ECGs will be obtained after the patient has been resting in a semi-recumbent position for at least 5 minutes. All digital ECGs will include the date and time obtained, heart rate, QRS duration, PR interval, RR interval, QT interval, and QTcF interval using Fridericia formula (Puddu et al., 1988). If indicated, additional ECG assessments may be performed, at the discretion of the investigator. If applicable, clinically significant changes from baseline in ECG assessments will be noted as AE(s), in accordance with Section 15.2.1.

# 15.7 Study Monitoring by the Drug Safety Monitoring Board (DSMB)

The study will be monitored for safety, futility, and efficacy by a DSMB. Interim analysis for safety will be conducted six weeks after the first 30-35 participants complete Day 42 based on reported Adverse Events and Serious Adverse Events. The study may be stopped for safety concerns. A second DSMB assessment for safety and futility will be conducted when 45-50 participants have reached day 42.

## 16. STATISTICS

The study analyses will be conducted in a GCP environment (ICH E6 and E9 [R1]). All analyses will be pre-specified in a Statistical Analysis (SAP) and finalized prior to database lock. If the methods in the SAP do not agree with this protocol, the methods described in the SAP will govern the analysis.

#### 16.1 Randomization

Randomization will be stratified by evidence of a suicidal event in the prior 12 months (none, any).

## 16.2 Study Populations

The study includes prospectively defined study populations. The Intent to Treat (ITT) population will include all participants who received at least one dose of the oral treatment and had any post–randomization efficacy assessments. The modified ITT (mITT) population will include the ITT population with at least one post-baseline efficacy observation; the mITT population will also exclude subjects with a major protocol deviation, e.g. ineligibility, unreliable MADRS-10 scoring, proscribed treatment. The Per Protocol (PP) population will include the subset of ITT participants who were eligible, who have any post–randomization efficacy assessments within one day of scheduled visits through Day 7 and within three days of scheduled visits through Day 42, and who had no major protocol violations. The Safety population will include all participants as treated with study treatment and with any post–randomization safety data.

The mITT population will be used for the primary analyses for efficacy. If <5 percent are to be excluded from the ITT population, then the analysis will not be performed for the PP population.

Protocol violations will be reviewed in real time and prospective rules will be set for exclusions from the PP population. A Biostatistics Data Review Meeting (BDRM) will be held to identify all major protocol deviations prior to database lock inclusive of any case exclusions from the mITT and PP population as well as to censor any efficacy data following proscribed treatments.

## 16.3 Hypothesis Tests

#### **16.3.1 Treatment Comparisons**

In order to preserve the Type 1 error associated with multiple endpoints (per FDA guidance), all efficacy endpoints will be evaluated in this pre-defined order: (1) MADRS through Week 6. Each will be hypothesis testing driven.

# 16.3.2 Primary Hypothesis

#### **MADRS**

The primary study hypothesis is that treatment with NRX-101 is superior to lurasidone in improving symptoms of depression as measured by the MADRS over 6 weeks of treatment. The primary study hypothesis is that treatment with NRX-101 is superior to lurasidone in improving

symptoms of depression as measured by the MADRS over 6 weeks of treatment. The null hypothesis for the primary endpoint is the mean change from baseline of MADRS-10 for NRX-101 is the same as lurasidone. Baseline is defined as MADRS-10 score at study entry.

The null hypothesis is no difference in the mean change in the MADRS-10 score from baseline to Day 42/exit between both treatment groups, while the alternative hypothesis is that there is a larger mean improvement in the NRX-101 group than the lurasidone group. The study is to have 80% power to detect a 0.66 effect size post-baseline for a two-sided test with 5% Type 1 error using mixed model repeated measures (MMRM).

# 16.3.3 Key Secondary Hypotheses

The key secondary hypothesis are that:

- treatment with NRX-101 is superior to lurasidone in improving symptoms of suicidality as measured by the CGI-SS over 6 weeks of treatment. The null hypothesis for the primary endpoint is the mean change from baseline of CGI-SS for NRX-101 is greater than or equal to the mean change from baseline of CGI-SS for lurasidone while the alternative hypothesis is that the mean change from baseline of CGI-SS is less than the mean change from baseline of CGI-SS for lurasidone (improvement). Baseline is defined as CGI-SS score at this study entry.
- that NRX-101 is superior to lurasidone in time to treatment failure as defined as: study discontinuation due to Adverse Events; psychiatric hospitalization; or requiring a change in antidepressant treatment. Time to treatment failure may be ascertained as the treating physician's determination of a study discontinuation due to lack of efficacy; withdrawal due to a treatment related adverse event a psychiatric hospitalization; or the patient requiring any change in their baseline antidepressant, mood stabilizer, or antipsychotic medication. Titration or change in timing of administration of study medication will not be considered a failure of therapy. Lack of efficacy is defined as the need to implement a new treatment plan or an increase in suicidal ideation (a score of 4 or 5 on the C-SSRS, emergent suicidality requiring hospitalization), or increase in depressive symptoms (a score increase of  $\geq$ 5 for two consecutive visits on the MADRS total score). The need to implement a new treatment plan includes the addition of new antidepressant medication or somatic treatment (e.g. ECT or rTMS treatment) or an escalation of care such as hospitalization (i.e. moving the patient from outpatient care to initiating inpatient, partial or day hospitalization). Time to failure will be assessed using a Kaplan-Meier lifetable. The formal hypothesis test will be to detect a 0.421 hazard ratio (HR) with 80% power for a two-sided test using a proportional hazard model; a 0.545 hazard ratio reaches two-sided p=0.05.

## 16.4 Efficacy Endpoints

# 16.4.1 Primary Efficacy Endpoints

The primary efficacy endpoint is the change from baseline in the total MADRS score as measured by psychometric raters assessed over 42 days post randomization by mixed-model repeated measures analysis.

# 16.4.2 Secondary Efficacy Endpoints

The key secondary efficacy endpoints are:

- Change from baseline in CGI-SS score as measured by treating prescriber assessed over 42 days post randomization by mixed-model repeated measures analysis.
- Time to Treatment Failure (TTF) A Kaplan-Meier lifetable will be constructed for the time to failure of therapy. Failure of therapy will be defined as the treating physician's determination of a study discontinuation due to lack of efficacy; withdrawal due to a treatment related adverse event a psychiatric hospitalization; or the patient requiring any change in their baseline antidepressant, mood stabilizer, or antipsychotic medication. Titration or change in timing of administration of study medication will not be considered a failure of therapy.

The additional efficacy endpoints are:

- Change from baseline to endpoint in Suicidal Thoughts on the MADRS (MADRS item 10)
- Mean change from baseline to Day 14 in total MADRS score
- Change from baseline to endpoint in each item of the Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 (clinical global impressions of frequency of suicidal thinking, severity of suicidality, and imminent and long-term risks)

# 16.4.3 Other Exploratory Efficacy Endpoints

The following other efficacy endpoints will be explored:

• Remission from suicidality: A Kaplan-Meier lifetable will be constructed for the remission duration from response onset where remission is defined as reaching CSSR-S ≤ 2 and remaining through the study. Remission rate is defined as percent remaining in remission.

Collectively, symptom improvement will be evaluated by assessing changes in the secondary outcome measures within and between treatment groups for each of the following at the times specified on the Schedule of Study Activities:

- Montgomery Asberg Depression Rating Scale (MADRS) (Montgomery, Åsberg 1979)
- Clinical Global Impression of Severity of Suicidality Scale (CGI-SS)

- Concise Health Risk Tracking Self Report (CHRT-SR) and Clinician Rating (CHRT-C) scales (Trivedi et al., 2011)
- Brief Psychiatric Rating Scale (BPRS) (Overall and Gorham, 1962).

# **16.4.4 Other Efficacy Endpoints of Interest**

The following additional endpoints will be recorded and analyzed by treatment group:

- Dose per treatment group
- Suicide rates (attempted and completed)
- Time to all-cause study discontinuation (and reason for discontinuation) due to any reason such as withdrawal due to an adverse event, or patient or investigator decision to withdraw
- Rate of participants who achieve a resolution of suicide risk by Clinical Global Judgement of Suicide Risk [CGI-SR] 0 or 1) or by MADRS (suicidal ideation item #10 of 0 or 1)
- Proportion of participants who are treated with new SSRIs or have increased SSRI dosages
- Proportion of participants who discontinue SSRIs or have reduced SSRI dosages
- Efficacy for each MADRS factor; mania, depression, irritability, anxiety, and psychosis

# 16.4.5 Diagnostic Metric

The following metrics will be evaluated at baseline:

• MINI 7.0.2

## 16.5 Safety Assessments

- Change from baseline to endpoint (Day 42) in C-SSRS score
- Change from baseline to endpoint (Day 14) in C-SSRS score
- Mean change in BARS through Day 42 to assess akathisia
- Percent in remission at Day 42/exit, defined as having achieved a MADRS score of ≤ 10 during the last two visits (14 days)
- Rates of discontinuation between the arms

#### **16.5.1 Overall Adverse Events**

Separate and combined safety analyses will be performed for the Safety population. All safety results will be presented separately for each treatment group. Safety endpoints will include adverse events (AEs), vital signs, ECGs, and laboratory parameters.

The principle of treatment emergence will be employed for the analysis of AE data. Treatment emergence is defined as any event that occurred following the initiation of therapy and was not

present at baseline, or one which represents an exacerbation of a condition present prior to study entry (pre-existing).

Unresolved AE outcomes at the end of the study will be followed for an additional seven days or until resolution, whichever occurs earlier.

Adverse events will be classified by the Medical Dictionary for Regulatory Activities (MedDRA). For each study treatment, safety data will be collected and analyzed until treatment-emergent AEs are resolved. The type, incidence, timing (onset, duration), relationship, and severity of treatment-emergent AEs will be reported. Reasons for withdrawal due to AEs will also be reported.

Two-sided Fisher Exact tests will be performed to compare the two treatment groups with respect to incidence at the system order class level and for any preferred terms with >10 percent overall incidence.

## 16.5.2 Other Safety Measures

The timing and incidence of adverse findings will be compiled following planned surveillance of all study participants by a designated safety monitor.

Vital signs and ECGs will also be evaluated within and between study treatment groups. The overall ECG interpretation will be reported as normal or abnormal; if abnormal, then the percent clinically significant will be reported.

While symptom improvement will be evaluated by assessing changes in the secondary outcome measures (CHRT, MADRS, and CGI-SS), safety measures in the C-SSRS, PRISE, BPRS, and BARS (including the global severity rating) will be evaluated within and between study treatment groups. The timeframe is for both lifetime and the past six months for the baseline Screening scale and since the last visit for the Since Last Visit scale.

## **16.6 Sample Size Calculations**

#### 16.6.1 Background

For DCS treatment group in major depressive disorder Heresco-Levy identified a 0.91 effect size for Hamilton-D Total and a 0.95 effect size for BDI-II (Heresco-Levy, 2013) and an effect size of >1 was seen in the phase 2 STABIL-B study with a similar effect size observed by Chen and Heresco-Levy.

A more modest 0.66 effect size is targeted in the sample size calculations assuming a 1:1 allocation for a two-sided hypothesis test with 5 percent Type I error.

## 16.6.2 Power and Significance

These sample size calculations are based on the alternative hypothesis corresponding to a 0.66 effect size which corresponds to a mean 8.85-unit MADRS-10 advantage change from baseline for NRX-101 vs control. A total of 74 subjects are to be randomized 1:1 to support the final analysis. As summarized below in Table 6, there is 80% power to detect a 0.66 effect size; a

0.462 effect size would reach two-sided p=0.05. A 0.462 (moderate) effect size reflects a 50 percent drop (based on lurasidone published data) in mean change from baseline for lurasidone with an assumed standard deviation of 13.4; this approximately corresponds to a -16 mean CFB for NRX-101 and a -10 mean CFB for lurasidone.

**Table 6** MADRS-10 Change From Baseline Outcomes: T-tests

| | Power | Significance |
|------------------------------------|-------|--------------|
| Test significance level, α | 0.05 | 0.05 |
| 1 or 2 sided test | 2 | 2 |
| Effect size, $d = m_1 - m_2 / s$ | 0.66 | 0.462 |
| Power (%) | 80 | NA |
| N per group | 37 | 37 |

The secondary efficacy hypotheses will also be evaluated using a hierarchical testing strategy where testing continues as long as two-sided p<0.05 is reached. The first such hypothesis to be tested will be for primary endpoint MADRS change from baseline to endpoint, then change from baseline in CGI-SS, followed by time to treatment failure in the NRX-101 and lurasidone groups.

# 16.6.3 Interim Analyses

Two interim analyses are planned. The first interim analysis (IA) assessing safety will be conducted six weeks after the first 30-35 participants have been followed for 6 weeks and the second IA assessing futility (primary efficacy endpoint) will be performed after the first 45-50 participants have been followed for 6 weeks.

Each interim analysis has a different objective with neither interim analysis spending any Type 1 error. The study will be stopped at the first interim analysis if Serious Adverse Events are deemed statistically significantly more common in the NRX-101 group compared to the lurasidone group in a manner deemed by the DMC to pose a potential danger to human subjects. The study will be stopped at the second IA for futility if the conditional power (CP) is less than 10%. In the event that the study is not stopped for either safety or futility, then enrollment will continue until a total of 74 subjects are randomized. This preserves two-sided p=0.05 for the final analysis.

The unblinded Sponsor biostatistician will perform the interim analyses for the Data Safety Monitoring Board (DSMB). The blinded Sponsor biostatistician will then adjudicate cases with respect to intercurrent events which impact analysis inclusion.

# 16.7 Adjudication of Primary Endpoint

All rating sessions for MADRS-10 and C-SSRS will be recorded as audio files and reviewed by central master-raters with > 25 years of experience. Any MADRS-10 total score the differs by more than three points from the master-rater score will be deemed non-congruent. All non-congruent subject-visits from any site with > 10% non-congruent scores will be sent to an independent adjudicator, previously determined to have > 90% concordance with study master

raters on standardized training data. In the event of adjudication as above, the independent outside rater score shall be considered as the subject-visit primary study endpoint.

#### 16.8 Statistical Analysis Approach

#### **16.8.1 Software**

All calculations will be performed using SAS statistical software, version 9.3 or later, and StatXact, version 10 or later.

## 16.8.2 Display Formats

All efficacy and safety data will be displayed in tables and listings separately for each treatment group.

#### 16.8.3 Conventions

Study visit dates will be analyzed using the nominal visit instead of the actual visit date.

Means, mean changes, standard deviations, and ranges will be presented separately for each treatment group. These endpoints will be evaluated using a paired t-test and between study treatment groups using an unpaired t-test at each time; these p-values will be presented as descriptive statistics.

For continuous variables, the mean, standard deviation, minimum, median and maximum will be presented, together with the total number of observations and the number of missing and non-missing values.

For ordinal and categorical variables, absolute and relative frequencies will be reported. Relative frequencies will be based on all observations and reported as percentages. Unless otherwise specified, percentages will be based on the number of participants with data and will not be calculated for missing categories.

Adverse events, medical histories, and concomitant medications will be reported on a patient and an event basis. Percentages will be calculated using the number of participants in the Safety population analysis set as the denominator.

All hypotheses will be tested at 5 percent (final analysis) level of significance using a two-sided test unless otherwise specified.

#### 16.8.4 Estimand Structure

Analyses will be conducted in accordance with ICH E9 (R1) analysis principles as summarized below.

| Primary scientific question of | The primary study hypothesis is that treatment with NRX- |
|---|---|
| interest | 101 is superior to lurasidone in improving symptoms of |
| | depression as measured by the MADRS over 6 weeks of |
| | treatment. The null hypothesis for the primary endpoint is |

| Target population | the mean change from baseline of MADRS-10 for NRX-101 is the same as lurasidone while the alternative hypothesis is that the mean change from baseline of MADRS-10 is larger than the mean change from baseline of MADRS-10 for lurasidone. Baseline is defined as MADRS-10 score at study entry. The mITT population will be the primary analysis population. The mITT population is defined through appropriate inclusion/exclusion criteria as specified in the |
|---|---|
| | protocol and blinded BDRM decisions. |
| Treatment of interest | NRX-101 |
| Outcome Variable | MADRS-10 (and C-SSRS) will be recorded as audio files and reviewed by central master-raters with any non-congruent subject-visits from any site with >10% non-congruent scores sent to a qualified independent adjudicator to be considered as the subject-visit primary study endpoint. |
| Summary Measure | The contrast-estimated MADRS-10 Week 6 MMRM will use all post-baseline data with LOCF in the mITT population excluding all outcomes after BDRM-approved exclusions. The model will include treatment and the following four baseline stratification factors in addition to baseline MADRS-10: (1) sex, (2) mood stabilizer use, (3) anti-psychotic use, and (4) evidence of suicide event in their lifetime. The model will include treatment group, study visit, the interaction between study visit and treatment group, baseline MADRS-10, and the four baseline covariates as fixed effects. An unstructured error structure will be assumed. |
| Intercurrent Events | A BDRM will adjudicate all intercurrent events which may redact outcomes after disqualifying events; these intercurrent events may represent major protocol deviations. Any ITT subject with no post-baseline MADRS-10 observations will use the baseline MADRS-10 observation to replace all post-baseline MADRS-10 observations. |

# 16.8.5 General Methodology

The Mixed-Effect Model Repeated Measure (MMRM) will be the primary analysis for the primary efficacy endpoint (MADRS change from baseline); an unpaired t-test will be a secondary analysis. The proportional hazard model (PHREG) will be the primary analysis for time to event endpoints (time to relapse, time to discontinuation); the unstratified log rank test will be a secondary analysis. The MMRM and PHREG models will all include treatment and the following four baseline stratification factors:

- sex
- mood stabilizer use
- anti-psychotic use
- evidence of suicide event in their lifetime.

All primary analyses will be in the ITT population as primary and repeated in the Per Protocol population if >5 percent are excluded.

All of the instruments used to measure SSIB or depression constitute serial continuous and ordinal outcomes that will be analyzed using MMRM with LOCF to account for missing data and early discontinuations. The models will include treatment group, study visit, the interaction between study visit and treatment group, the baseline level of the variable being analyzed, and the above four pre-defined baseline stratification factors as fixed effects. The primary endpoint change from baseline MADRS-10 will be analyzed using the MMRM model which will include baseline MADRS; treatment group; study visit; study visit\*treatment; sex, mood stabilizer use, antipsychotic use, and evidence of suicide event in their lifetime as defined above. An unstructured error structure will be assumed.

SAS PROC MIXED will be used for continuous endpoints and PROC GENMOD will be used for binary endpoints.

In addition, multiple imputation will be performed to address any missing data. The method of Little and Rubin will be used. The presentation of the results for the primary efficacy endpoints using the ITT population will be based on the observed data with multiple imputation for missing endpoint data using SAS PROC MI. Missing data will be imputed using MCMC imputation under the assumption of a missing at random using the ITT population. The SAS® procedure PROC MI will be used for the MCMC imputation of 25 complete data sets.

#### **16.8.6** Other Time to Event Efficacy Endpoints

Other time-to-event outcomes (all-cause discontinuation, and remission duration) further characterize this multi-component disorder. Time to event is a more sensitive measure than an assessment at a fixed time. Time to such events will be displayed using a Kaplan-Meier lifetable, with the treatment groups compared using two-sided unstratified log rank tests (secondary) and a proportional hazard model (primary) to include the above cited baseline covariates.

Treatment Failure will be centrally judged blind in real time by the study physician using baseline measures of depression and suicidality as a guide. Treatment failure is defined above.

# 16.8.7 Secondary Efficacy Endpoints

All of the instruments used to measure SSIB or depression constitute serial continuous and ordinal outcomes that will be analyzed using MMRM with LOCF, which accounts for missing data and early discontinuations. Results will be presented separately for each treatment group.

The models will include treatment group, study visit, the interaction between study visit and treatment group, the randomization baseline of the variable being analyzed, and the three baseline stratification factors as fixed effects. The reason for missing data will be evaluated as a condition of MMRM analysis.

## 16.8.8 Other Endpoints of Interest

The following additional endpoints will be recorded and analyzed by treatment group for both study phases:

- Dose per treatment group
- Suicide rates
- Proportion of participants who are treated with new SSRIs or have increased SSRI dosages
- Proportion of participants who discontinue SSRIs or have reduced SSRI dosages
- Efficacy for each BPI factor.

Dose per treatment group will be displayed graphically over time per study treatment group. The percent decreasing and increasing over time relative to starting dose will be displayed per study treatment group.

Time to all-cause study discontinuation and time to discharge will be displayed using a Kaplan-Meier lifetable.

The following three measures will be separately evaluated using a two-sided Fisher Exact test to compare treatments:

- the need to implement a new treatment plan.
- an increase in suicidal ideation (a score of  $\geq 4$  on the C-SSRS, emergent suicidality requiring hospitalization).
- an increase in depressive symptoms (a score increase of  $\geq 5$  for two consecutive visits on the MADRS total score).

The incidence of hospitalization and ER visits will be evaluated using a Wilcoxon Rank Sum test to compare each study treatment group.

The proportions of participants discontinuing SSRIs or reducing SSRI dosages will be displayed graphically over time per study treatment group. The percent discontinuing SSRIs and reducing SSRI dosages relative to starting dose will be displayed per study treatment group.

# 16.8.9 Safety Endpoints

Adverse events will be classified by MedDRA. For each study treatment, safety data will be collected and analyzed while on treatment or until treatment-emergent adverse events are resolved. The type, incidence, timing (onset, duration), relationship, and severity of AEs will be reported for treatment-emergent and SAEs. Reasons for withdrawal due to AEs will also be reported. Narratives will be written for every AE classified as serious or associated with attempted suicide or death.

Safety and tolerability will be assessed using two-sided Fisher Exact tests to compare overall adverse event incidence for NRX-101 vs. lurasidone. Mean changes from randomization baseline will be displayed for each serum chemistry and hematology parameter as well as the shift; unpaired t-tests will be used to compare treatments. In addition, paired t-tests will be performed for the changes from randomization baseline for each study treatment group.

Vital signs and ECGs (means and mean changes from baseline will also be evaluated within treatment groups using paired t-tests and between study treatment groups using unpaired t-tests. Percent with abnormal vital signs, heart rate, QRS duration, PR interval, RR interval, QT, and QTcF will be reported. McNemar paired comparison tests will be performed within study treatment groups for the abnormal discordant percent while two-sided Fisher Exact tests will be performed to compare incidences between treatment groups.

Blood draws for chemistries and hematologies will be evaluated within and between study treatment groups. Abnormality rates will be presented relative to established site-specific normal ranges and whether or not the abnormality is clinically significant. McNemar paired comparison tests will be performed within study treatment groups for the abnormal percents while two-sided Fisher Exact tests will be performed to compare incidences between treatment groups.

#### 17. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 17.1 Study Monitoring

Potential study sites will be evaluated by the sponsor in conjunction with the CRO to determine suitability for the proposed study. Information reviewed will include, but will not be limited to, facility details and site capabilities, past performance in similar studies, investigator and staff experience, ongoing studies at the site, projected enrollment, and FDA or other agency audit findings. Study sites may be asked to complete a study-specific Site Selection Questionnaire and other documents for consideration for participation, and clinical study monitors may make a Site Qualification Visit prior to completing the evaluation process. Upon completion of this evaluation, the sponsor will invite the chosen sites for participation.

Prior to patient enrollment, a study initiation visit will be completed at each investigational site to ensure the following: IRB approval has been obtained and documented prior to patient screening, the investigators and study personnel are appropriately trained and clearly understand the study, and the investigators and study personnel accept the obligations incurred in undertaking this clinical investigation. Due to the current COVID-19 Pandemic these visits may be a virtual videoconference visit.

Raters proposed by each site will be evaluated on the basis of experience and education for each instrument used in the study. Raters with the appropriate levels of experience and education will be trained by an independent third party in the use of each instrument and approved to administer that instrument in the study. Sites will not be approved to begin enrollment activities until they have at least one rater approved for each clinician-administered instrument (See Appendix 3: Rater Training Manual).

Qualified clinical monitors will conduct investigational site monitoring visits on a routine basis to ensure that all investigators conduct the study in compliance with the protocol and applicable regulations. These monitoring visits may be virtual visits video/teleconference visits. The site will receive notification prior to each monitoring visit during the course of the study. It is expected that the investigator and/or sub-investigator and other appropriately trained study staff are available on the day of the visit in case any questions may arise. Due to the Pandemic situation, sites may also provide a secure access to portions of electronic medical records, and or upload de-identified information onto a secure platform.

Periodic monitoring visits will be made in accordance with the approved monitoring plan at all active study sites throughout the clinical study to ensure that the investigator obligations are being fulfilled and all applicable regulations and guidelines are being followed. These visits will assess continued acceptability of the facilities, ensure the protocol and investigational plan are being followed, the IRB has been notified of approved protocol changes as required, complete records are being maintained, appropriate and timely reports have been made to the sponsor, CRO, and the IRB, and the site's Principal Investigator is executing all agreed activities.

The sponsor retains the right to remove either the Principal Investigator or the investigational site from the study for issues of non-compliance with the protocol or regulatory requirements.

On one or more occasion, the study site may be inspected or audited by the sponsor representative or a third party. The investigator will be informed in advance of the visit(s).

Upon completion of the clinical study (when all participants at the site have completed follow up visits, all data has been entered in EDC and cleaned, all queries resolved, and final electronic signatures have been obtained), a study closeout visit will be performed. Any unused study materials and equipment will be collected and returned to the depot. The monitor will help to ensure that the investigator's regulatory files are up to date and complete and that any outstanding issues from previous visits have been resolved. Other issues that will be reviewed at this visit

include: discussing retention of study files, possibility of site audits, publication policy, and ensuring that the investigator will notify the IRB regarding study closeout.

#### 17.2 Audits and Inspections

The Sponsor and its representatives will have direct access to source data and documents for study monitoring. Additionally, the IRB and FDA may review source data following appropriate guidelines for this process.

#### 17.3 Institutional Review Board (IRB)

The study protocol and any amendments will be reviewed by an IRB. The IRB will review the informed consent form, their updates (if any), and any written materials given to the participants.

IRB approval will be obtained and documented prior to patient enrollment and screening. Before study initiation, the investigator must have written and dated approval from the IRB for the protocol, consent form, patient recruitment materials/process (e.g., advertisements), and any other written information to be provided to participants.

The investigator will provide the IRB with reports, updates, and other information (e.g., Safety Updates, Amendments, and Administrative Letters) according to regulatory requirements and Institution procedures.

A detailed list of required regulatory documents to be submitted to the CRO and/or sponsor, will be sent upon final approval of the protocol.

# 18. QUALITY CONTROL AND QUALITY ASSURANCE

#### 18.1 Source Data and Records

Source data are all the information in original records and certified copies of original records of clinical findings, observations, laboratory reports, and data sheets provided by the sponsor or other activities in the study, that are necessary for the reconstruction and evaluation of the study. The investigator will permit study-related monitoring, audit(s), IRB review(s), and regulatory inspection(s), with direct access to all the required source records.

All study records will be retained for at least two years following the date on which the drug is approved by the regulatory authority for marketing for the purposes that were the subject of the investigation. In other situations (e.g., where the investigation is not in support of or as part of an application for a research or marketing permit), the requirement will be two years following the date on which the entire clinical program is completed, terminated, or discontinued, or when the investigational application under which the investigation is being conducted is terminated or withdrawn by the regulatory authorities.

In the event the site's Principal Investigator retires, relocates or for any other reason withdraws from the responsibility for maintaining records for the period of time required, custody of the records may be transferred to any other person who will accept responsibility for the records. Notice of such a transfer must be given in writing to the Sponsor. The Investigator must contact the Sponsor prior to disposal of any records related to this study.

## 18.2 Reporting Study Data

The eCRF is an integral part of the study and subsequent reports. The eCRF will be used to capture all study data recorded in the patient's medical record that is applicable to this study. The eCRF must be kept current to reflect patient status during the course of the study.

All protocol-required information collected during the study must be entered by the Investigator, or designated representative, in the eCRF, an Internet-based electronic data collection system. All details regarding eCRF completion and correction will be explained to the investigator. The eCRF includes edit check and query systems that seamlessly integrate with the data entry system. All modifications to the data in the eCRF are tracked by an electronic audit trail (date and identity of the person making the change are instantaneously recorded). The eCRF is 21CFR Part 11 compliant.

If the investigator authorizes other persons to make entries in the eCRF, the names, positions, and signatures of these persons must be supplied to the sponsor.

The Investigator, or designated representative, should complete the eCRF as soon as possible after information is collected, preferably on the same day that a study patient is seen for an examination, treatment, or any other study procedure. By design, an explanation must be provided for all missing data, altered data, and/or out of range data.

The completed eCRF must be reviewed and signed by the site's Principal Investigator or by a designated sub-investigator.

Final monitored eCRFs will be provided by the sponsor to the sites at the end of the study in the format of a PDF file for archival purposes.

# **18.2.1** Clinical Trial Registry

The study will be posted to Clinicaltrials.gov, and results will be reported in accordance with Clinicaltrials.gov guidelines.

#### 18.3 Confidentiality of Patient Data

The risk of loss of privacy is judged to be minimal. Sites will enter patient data directly into the eCRF, which will be managed by the CRO or contracted data management company. Participants will be assigned study ID numbers.

Potential risks to data confidentiality will be mitigated by requirements for the de-identification of all study data and by security protocols for all data capture systems. All users will be tracked and

NRX-101 003  09 NOVEMBER 2023

provided access in a secure fashion following established Standard Operating Procedures (SOPs) for this process.

As with all research data, information gathered by the study will be used only for aggregate analysis; it will not be released with any information that identifies research participants. Uses and risks related to data collection will be outlined in the informed consent and reviewed with the participants.

# 19. ETHICAL CONSIDERATIONS

## 19.1 Ethical Conduct of the Study

This study will be conducted in accordance with the ethical principles that have their origins in the Declaration of Helsinki, in compliance with the approved protocol, GCP, and applicable regulatory requirements.

Participants must be capable of understanding the nature of this study, its potential risks, discomforts, and benefits. Study physicians will obtain consent after they have fully explained the study purpose and its procedures, and after potential participants have demonstrated an understanding of the protocol, willingness to participate, and competency to consent.

#### 19.2 Patient Information and Consent

Participants must be capable of understanding the nature of this study and its potential risks, discomforts, and benefits. Study physicians will obtain consent after they fully explain the study purpose and its procedures, and the potential patient demonstrates an understanding of the protocol, willingness to participate, and competency to consent.

The investigator must ensure that participants are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical trials in which they volunteer to participate. Preparation of the site-specific informed consent form is the responsibility of the site Principal investigator and must include all elements required by CFR 21 Part 50.25 and the IRB.

Each patient will receive the informed consent form for the study. The document will be read by the patient and also reviewed by the patient with a clinician on the research staff prior to participating in the study. Any questions, concerns, or ambiguities will be clarified by the site investigator or another study clinician prior to the patient signing the informed consent form. Participants will only begin study participation after signing the informed consent form.

# 20. REFERENCES

- Aiken, C.B., Weisler, R.H., & Sachs, G.S. (2015). The Bipolarity index: a clinician-rated measure of diagnostic confidence. *Journal of Affective Disorders*, 177, 59–64.
- Alphs L, Canuso C, Williamson D. P.1.k.032 The Suicide Ideation and Behavior Assessment Tool: development of a novel measure of suicidal ideation and behavior and perceived risk of suicide. *Eur Neuropsychopharmacol*. 2015;25:S371.
- Barnes TR. A rating scale for drug-induced akathisia. Br J Psychiatry. 1989 May;154:672-6
- Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, et al. Antidepressant effects of ketamine in depressed patients. Biol Psychiat. 2000;47(4):351-4.
- Coryell W, Kriener A, Butcher B, Nurnberger J, McMahon F, Berrettini W, Fiedorowicz J. Risk factors for suicide in bipolar I disorder in two prospectively studied cohorts. J Affective Disorders. 2016; 190:1-5.
- Crane GE. Cycloserine as an anti-depressant agent. Am J Psychiat. 1959;115:1025–9.
- Crane GE. The psychotropic effects of cycloserine: a new use for an antibiotic. Compr Psychiat. 1961;2:51–9.
- Cyrus R. Mehta, Stuart J., Pocock. Adaptive Increase in Sample Size when Interim Results are Promising: A Practical Guide with Examples. Statist. Med. 2000; 00:1–6.
- Harada T, Inada K, Yamada K, Sakamoto K, Ishigooka J. A prospective naturalistic study of antidepressant-induced jitteriness/anxiety syndrome. Neuropsychiatric disease and treatment. 2014;10:2115-21.
- Heresco-Levy U, Javitt DC, Gelfin Y, Gorelik E, Bar M, Blanaru M, et al. Controlled trial of D-cycloserine adjuvant therapy for treatment-resistant major depressive disorder. J Affect Disorders. 2006;93(1-3):239-43.
- Heresco-Levy U, Gelfin G, Bloch B, Levin R, Edelman S, Javitt DC, et al. A randomized add-on trial of high-dose D-cycloserine for treatment-resistant depression. Int J Neuropsychop. 2013;16(3):501-6.
- Hood WF, Compton RP, Monahan JB. D-cycloserine: a ligand for the N-methyl-D-aspartate coupled glycine receptor has partial agonist characteristics. Neurosci Lett. 1989;98(1):91-5.
- Javitt DC, Composition and method for treatment of psychosis and depression in humans. US patent application 2014/0018348, filed Jan 2014. www.uspto.gov.
- Javitt D, Nirenberg A, Mathew S, et. al. Sequential Treatment With IV Ketamine Followed by Combined Oral D-Cycloserine + Lurasidone (NRX-101) forSevere Bipolar Depression and Suicidality: Preclinical and Clinical Findings. Neuropsychopharmacol 2018:W134. https://doi.org/10.1038/s41386-018-0268-5

- Kessler RC, Chiu WT, Demler O, Walters EE. Prevalence, severity, and comorbidity of twelvemonth DSM-IV disorders in the National Comorbidity Survey Replication (NCS-R). Archives of Genera. Psychiatry, 2005 Jun;62(6):617–27.
- Krystal JH, Bennett A, Abi-Saab D, et al. Dissociation of ketamine effects on rule acquisition and rule implementation: possible relevance to NMDA receptor contributions to executive cognitive functions. *Biol Psychiatry*. 2000;47(2):137–43.
- Little R, Rubin D. Statistical Analysis with Missing Data. John Wiley and Sons, New York 2002.
- Loebel A, Cucchiaro J, Silva R, Kroger H, Hsu J, Sarma K, et al. Lurasidone monotherapy in the treatment of bipolar I depression: a randomized, double-blind, placebo-controlled study. Am J Psychiat. 2014a;171(2):160–8.
- Loebel A, Cucchiaro J, Silva R, Kroger H, Sarma K, Xu J, et al. Lurasidone as adjunctive therapy with lithium or valproate for the treatment of bipolar I depression: a randomized, double-blind, placebo-controlled study. Am J Psychiat. 2014b;171(2):169–77.
- Lopes T, Neubauer P, Boje KM. Chronic administration of NMDA glycine partial agonists induces tolerance in the Porsolt swim test. Be. 1997;58(4):1059–64.
- Mahli, GS, Thoughts on suicidal thinking in bipolar disorder. Bipolar Disord. 2015 Feb; 17(1):19–21. doi: 10.1111/bdi.12276. Epub 2014 Nov 3.
- Mehta CR, Pocock SJ. Adaptive Increase in Sample Size when Interim Results are Promising: A Practical Guide with Examples. Statist. Med. 2011; 30, 28, 3267-3284.
- Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Brit J Psychiatry 1979;134(4):382-89.
- Nierenberg, A. A., Gray, S. M., & Grandin, L. D. (2001). Mood disorders and suicide. *J Clin Psychiatry*, 62 Suppl 25, 27-30.
- Overall JE, Gorham DR. The Brief Psychiatric Rating Scale. *Psychol Rep.* 1962;10(3):799-812.
- Pompili M, Gonda X Serafini G. Epidemiology of Suicide in Bipolar Depression. Bipolar Disorders. 2013;15(5):457-90.
- Popovic D, Vieta E, Azorin JM, Angst J, Bowden CL, Mosolov S, et al. Suicide attempts in major depressive episode: evidence from the BRIDGE-II-Mix study. Bipolar Disorders. 2015.
- Posner K, Oquendo MA, Gould M, Stanley B, and Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry 2007. 164:1035-43.
- Puddu PE., Jouve R., Marlotti S., et al. Evaluation of 10 QT prediction formulas in 881 middle-aged men from the Seven Countries study: emphasis on the cubic root Fridericia's equation. J Electrocardiol 1988. 2:219–29.

- Rush, A.J., Asberg, M., 1999. Patient Rated Inventory of Side Effects (PRISE). Unpublished rating scale. University of Texas, University of Texas Southwestern Medical Center, Dallas.
- Sachdev PS, Brune M. Animal models of acute drug-induced akathisia a review. Neurosci Behav R. 2000;24(3):269–77.
- Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, et al. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59:22–33.
- Skolnick P, Layer RT, Popik P, Nowak G, Paul IA, Trullas R. Adaptation of N-methyl-D-aspartate (NMDA) receptors following antidepressant treatment: implications for the pharmacotherapy of depression. Pharmacopsychiatry. 1996;29(1):23-6.
- Stone M, Laughren T, Jones ML, Levenson M, Holland PC, Hughes A, et al. Risk of suicidality in clinical trials of antidepressants in adults: analysis of proprietary data submitted to US Food and Drug Administration. BMJ. 2009;339: b2880.
- Tan XL, Kern DM, Cepeda MS. Identifying Anticipated Events of Future Clinical Trials by Leveraging Data from the Placebo Arms of Completed Trials. Ther Innov Regul Sci. 2021 Mar;55(2):454-461. doi: 10.1007/s43441-020-00237-w. Epub 2020 Nov 9. PMID: 33165761; PMCID: PMC7864837.
- Targum SD, Pendergrass JC. Site-independent confirmation of subject selection for CNS trials: 'dual' review using audio-digital recordings. *Ann Gen Psychiatry*. 2014;13(1):21.
- Trivedi MH, Wisniewski SR, Morris DW, Fava M, Gollan JK, Warden D, Nierenberg AA, Gaynes BN, Husain MM, Luther JF, Zisook S, Rush AJ Concise Health Risk Tracking scale: a brief self-report and clinician rating of suicidal risk J Clin Psychiatry 2011 Jun 72 6 757-64.
- Trullas R, Skolnick P. Functional antagonists at the NMDA receptor complex exhibit antidepressant actions. Eur J Pharmacol. 1990;185(1):1-10.
- Wisniewski SR, Rush AJ, Balasubramani GK, Trivedi MH, Nierenberg AA, for the STARD Investigators. Self-rated global measure of the frequency, intensity, and burden of side effects. J Psychiatr Pract 2006;12:71–9.

# 21. APPENDICES

Appendix 1: Concomitant Medications

Appendix 2: Assessment Tools (provided as separate document)

Appendix 3: Rater Training Manual

Appendix 4: Medications Indicated for Use in Bipolar Disorder

NRX-101\_003  09 NOVEMBER 2023

# **Appendix 1** Concomitant Medications

Medications Allowed (Y) and Not Allowed (N) as Concomitant Medications

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Analgesics | Y | Y | Nonnarcotic analgesics are allowed. Medically appropriate episodic use of narcotic analgesics is allowed for acute medical indications but is limited to no more than three days for each episode. Chronic NSAID use is exclusionary; tramadol is also not allowed. |
| Anesthetics, general | Y<br>(except for<br>ketamine,<br>which is<br>excluded) | | If procedures requiring general anesthesia are to occur/have occurred, please contact Medical Monitor to report the medical condition(s). |
| Anesthetics, local | Y | N | _ |
| Anorexics | N | N | _ |
| Antacids | Y | Y | _ |
| Antiacne | Y | Y | Topical agents only, including topical antibiotics. Isotretinoin (Accutane) is not allowed. |
| Antianginal agents | N | N | _ |
| Antiarrhythmics | N | N | Amiodarone is excluded. |
| Antiasthma agents | Y | Y | _ |
| Antibiotics | Y | Y | Chronic use of topical antibiotics for acne is allowed, with the exception of the MAOI linezolid (Zyvox) and isoniazid, which are not allowed. Nafcillin, Erythromycin, clarithromycin, rifampin are excluded. |
| Anticoagulants | N | N | Warfarin (Coumadin) is not allowed. Antiplatelet agents are allowed (see "Antiplatelets"). |
| Anticholinergics | Y | Y | Except for scopolamine. |
| Anticonvulsants | N | Y | Gabapentin, lamotrigine and pregabalin are allowed. Other anticonvulsants are not allowed, including carbamazepine and oxcarbamazepine, phenytoin, phenobarbital, rufinamide (CYP3A4 inducers). Stable in dosing at least four weeks prior to randomization is required. |

NRX-101\_003  09 NOVEMBER 2023

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Antidepressants | N | Y | Stable (for at least 4 weeks prior to screening), ongoing antidepressant therapy is required during the course of the study. No dose changes are allowed during the study. Monoamine oxidase inhibitors (which may have unknown drug-drug interactions) are excluded. Concomitant use of trazodone (up to 200mg daily) is allowed. Nefazodone and St John's Wort are excluded (CYP3A4 inhibitor, inducer, respectively). |
| Antidiarrheal preparations | Y | | Only loperamide HCl (Imodium), bismuth subsalicylate (Pepto-Bismol), and kaolin preparations are allowed. |
| Antifungals, systemic | N | | Ketoconazole, itraconazol, rifampin and rifabutin are excluded. |
| Antifungals, topical | Y | Y | Ketoconazole and itraconzole are excluded. |
| Antihistamines | Y | Y | The use of combinations containing pseudoephedrine or phenylephrine is not allowed. Combination products containing the word nighttime or are specifically marketed for before sleep routinely include an antihistamine and are not allowed. Combination products ending in "-D" routinely contain a stimulant such as phenylephrine, and the appropriate limits above apply to them. (See "Cough and Cold Preparations" for combination products.) |
| Antihypertensives | N | Y | Diltiazem, verapamil are excluded. |
| Anti-impotence medications | Y | Y | _ |
| Anti-inflammatory drugs | Y | Y <sup>a</sup> | Indomethacin (Indocin) and systemic corticosteroids are not allowed. Chronic NSAID use is exclusionary. |
| Antimigraine | N | N | Triptans are not allowed. |
| Antinauseants/<br>Antiemetics | Y | | Phosphoric acid preparations (Emetrol, Emecheck), bismuth subsalicylate (Pepto-Bismol), cola syrup, 5-HT <sub>3</sub> receptor antagonis (e.g., ondansetron), and prokinetic agents (metoclopramide) are allowed. Scopolamine is not allowed (see section on anticholinergic). |
| Antineoplastics/<br>Immunosuppressant agents | N | Y <sup>c</sup> | Interferons, methotrexate, and other immunosuppressant agents are not allowed. Call Medical Monitor for approval for certain cases in cancer remission maintaining therapy. |

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Antiobesity/Appetite suppressants | N | N | OTC Alli (Xenical), sibutramine (Meridia), and phentermine (Adipex-P and others) are not allowed. |
| Antiplatelet agents | N | Y <sup>b</sup> | Aspirin (maximum 325 mg/day) and clopidogrel (Plavix) are allowed. Note that use of an SSRI or of a triple uptake inhibitor may increase bleeding times and possibly prothrombin times. |
| Antipsoriatic treatments | Y | Y | Only topical agents are allowed. Acitretin (Soriatane) is not allowed. |
| Antipsychotics | N | Y | Stable in dosing at least four weeks prior to randomization is allowed. Lurasidone will be discontinued at study entry. Quetiapine, aripiprazole, risperidone, brexpiprazole, olanzapine, cariprazine, or lumateperone should be discontinued prior to randomization. |
| Antismoking medications | N | Y <sup>c</sup> | Varenicline (Chantix) is not allowed. Chronic nicotine replacement may be allowed in certain cases after review with Medical Monitor. |
| Antiviral agents | Y | Y | Only oral or topical agents are allowed. Only acyclovir, famciclovir, valacyclovir, penciclovir, docosanal, trifluridine, and vidarabine are allowed. Amantadine, rimantadine, and protease inhbitors (atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir) are not allowed. Tamiflu (oseltamivir phosphate), and Relenza (zanamivir) inhalants are permitted for influenza prophylaxis but use is limited to a 7- to 14-day course in accordance with prescribing information. Interferons are not allowed. |
| Anxiolytics | N | Y | Chronic, stable treatment with benzodiazepines is allowed. Stable in dosing at least four weeks prior to randomization is required. |
| Barbiturates | N | N | Barbiturates are not allowed. |
| Benign prostatic<br>hyperplasia treatments | N | Y <sup>b</sup> | Male patients who have symptoms of obstructed voiding should not be included in the study. Surgically or medically treated patients must be asymptomatic and receiving a stable dosage of allowed medications (α-1 blockers, finasteride, or dutasteride) for one month before screening. |
| Buspirone | N | Y | Stable in dosing at least four weeks prior to randomization is allowed. |

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Cough/cold preparations | Y | N | Use of cough and cold preparations containing pseudoephedrine or dextromethorphan is not allowed, as are those containing phenylephrine Combination products ending in "-D" routinely contain a stimulant such as phenylephrine, and the appropriate limits apply to them. (See "Antihistamines".) |
| Diuretics | Y | Y <sup>b</sup> | Episodic use of diuretics is restricted to treatment of premenstrual symptoms. For chronic use, medication and dosage should be stable for 1 month before screening. |
| Dopaminergics | N | Y | Dopamine agonists for restless leg syndrome are allowed. |
| Ethyl alcohol | N | N | Participants should not use alcohol during the course of the trial because ethyl alcohol may increase the possibility and risks of seizures in participants receiving cycloserine. |
| Gastrointestinal: • H <sub>2</sub> -blockers/ • proton pump inhibitors/ • prokinetic agents | Y | Y | Cimetidine (Tagamet) is not allowed.<br>Metoclopramide is not allowed. |
| Hormonal (noncontraceptive) therapies | N | Y | See below. |
| Hormone suppressants | N | Y <sup>b</sup> | Only finasteride (Proscar) and dutasteride (Avodart) are allowed. |
| Hormones: reproductive | N | Y | Systemic hormonal contraceptives (oral contraceptives of estrogen and progestin combinations, depot injections such as Depo-Provera, the contraceptive implant Implanon, and/or transdermally delivered contraceptives such as Ortho Evra) are allowed. |
| Hormones: thyroid | N | Y | Thyroid hormone replacement is allowed (dosage of thyroid medication should be stable for three months before screening). Therapeutic use for psychiatric disorders (e.g., T3 augmentation) is not allowed. |
| Hypoglycemic agents | N | Y | Oral hypoglycemic agents are allowed. Insulin is allowed. |
| Hypolipidemics | N | Y <sup>b</sup> | Ezetimibe (Zetia) is allowed. |

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Hypolipidemics:<br>bile acid sequestrants | N | N | _ |
| Hypolipidemics: fibrates | N | Y <sup>b</sup> | Gemfibrozil and fenofibrate are allowed |
| Hypolipidemics: niacin | N | N | Niacin and niacinamide are not allowed. |
| Hypolipidemics: statins | N | $Y^b$ | Lovastatin, simvastatin, pravastatin, atorvastatin, fluvastatin, and rosuvastatin are allowed. |
| Laxatives | Y | Y <sup>a</sup> | Only fiber-based products and docusate sodium (Colace) are allowed. |
| Lithium | N | Y | Stable in dosing at least four weeks prior to randomization is allowed. |
| Medications that are primarily metabolized by CYP2C8 (e.g., cerivastatin, paclitaxel, repaglinide, sorafenib, and torsemide) | N | N | |
| Muscle relaxants | N | N | _ |
| NMDA receptor antagonist | N | N | Memantine is excluded. |
| Opioid agonists/analgesics (e.g., codeine, hydrocodone, methadone, morphine, maperidine, propoxyphene) and antagonists (e.g., naltrexone, naloxone, nalmefene) | N* | N* | See section on analgesics for exceptions. |
| Sedatives/hypnotics | N | | Ongoing, stable hypnotic therapy (e.g., zolpidem, zaleplon, benzodiazepine hypnotics, and low-dose trazodone 50-200mg) will be allowed during the course of the study. Eszopiclone is not allowed. |
| Steroids/systemic | Y | | Systemic steroid treatment will be allowed only for medical emergencies, such as severe allergic reactions. |
| Steroids/topical and inhalant | Y | Y | |
| Steroids/intra-articular | Y | NA | _ |

| Drug Name or Class | Episodic Use<br>(PRN) | Chronic Use | Restrictions/Comments |
|---|---|---|---|
| Stimulants | N | N | Oral or transdermal methylphenidate,<br>amphetamine products or prodrugs,<br>pseudoephedrine, modafinil (Provigil), and other<br>medications of same category are not allowed. |
| Vaccines | Y | NA | _ |

- a If being taken prior to enrolling in the study.
- b If being taken for at least three months prior to enrolling in the study and the dose has been stable for at least 1 month.
- c If approved by Medical Monitor5-HT<sub>3</sub> = 5-hydroxytryptomine receptor type 3; 5-HTP = 5-hydroxytryptophan; ACE = angiotensin-converting enzyme; CR = controlled release; DHEA = dehydroepiandrosterone; N = no; NA = not applicable; OTC = over the counter; PRN = as needed (prorenataT3prorenataT3=triiodothyronine; Y = yes.

NRX-101\_003  09 NOVEMBER 2023

# **Appendix 2** Assessment Tools

(Provided as separate document)

- MINI (version 7.0.2)
- C-SSRS (and the retrospective C-CASA component)
- CHRT (CHRT-SR and CHRT-C)
- MADRS
- PRISE
- CGI-Severity Suicidality (SIBAT Module 7)
- BPRS-psychosis subscale
- BARS

# **Appendix 3** Rater Manual: Rater Training & Certification Documentation

STANDARD OPERATING POLICY AND PROCEDURE FOR NRX RATER TRAINING & CERTIFICATION DOCUMENTATION

SOP General\_001-V1 Issue Date: 27-Feb-2023 Effective Date: 01-MAY-2019 Author: Marc Korczykowski

RATER TRAINING & CERTIFICATION DOCUMENTATION

Supersedes Document: 17Sept 2019

#### 1. POLICY

To establish NRX Policy for psychometric Rater Training that adheres to site level Institutional and Federal Regulatory Guidelines. This Policy is central to the protection of human subjects participating in research-related activities and extends to all NRX Staff, <<CRO or Designees, including Prevail Infoworks, Obvio Health, etc>> engaged in Clinical Trial activity. All Training, Certification, and documentation activity will be designed, implemented, and overseen by NRX Rater Program Manager, working in concert with Clinical Operations and Regulatory Affairs, which will review and approve all related processes, guidelines, and documentation *in compliance with NRX and Federal Regulatory Guidelines*.

#### 2. SCOPE

The scope of this Policy applies to all studies conducted by NRX, and is summarized in the NRX Rater Training Guidelines [V4] and NRX 101-003 Psychometric Rater Training 22Aug22 V5 documents. These policies and procedures apply to NRX, its employees, <<CRO or Designees, including Prevail Infoworks, Obvio Health, etc >> as well as subcontractors and others who train, manage, oversee and conduct research regulated by the FDA. Rater Experience Surveys will document that Staff performing study procedures are appropriately trained. Further, protocol-specific Psychometric Rater Training will also be completed prior to the initiation of the study-specific assessments. All Documentation and Training will be updated during the study if there are any changes to the personnel completing psychometric assessments. All Rater Training documentation will be maintained by the NRX Rater Program Manager, and copies will be shared with the <<CRO or Designees, including Prevail Infoworks>> Trial Master File for Study Documentation purposes. The scope of procedures applies to all clinical trial related psychometric assessments, including planning, performing data collection and reporting the results. Rater Training will be overseen by NRX Rater Program Manager, working in concert with <<CRO or Designees, including Prevail Infoworks>> and the Site Principal Investigator, who will supervise site level Psychometricians and Study Coordinators.

#### 3. RESPONSIBILITY

NRX and the Site Principal Investigator share responsibility for ensuring that all Psychometricians are qualified by training and experience to conduct their designated research-related duties. The NRX Rater Program Manager is responsible for providing initial and continuing training to all personnel, documenting and filing training certifications accordingly, and assessing training effectiveness through appropriate testing strategies. The NRX Rater Program Manager will ensure that protocol-specific psychometric assessments will be completed by an individual who has

NRX-101 003  09 NOVEMBER 2023

achieved the necessary education, experience, qualifications, and protocol-specific training to complete study-specific psychometric assessments. The Rater Program Manager will also implement training effectiveness measures for primary and secondary clinical endpoints. All Rater Training records will be signed by the both the Rater Program Manager and Study Staff member receiving the training. Training will reflect both General and Study-Specific conduct of psychometric assessments for human subjects research. The **Rater Qualification Approval Form** will be completed and signed by the Rater Program Manager when all training is complete. Training, including HIPAA & GCP certifications, will be maintained in the General and Study-Specific Regulatory Binders (e.g. eMSB or EDC), and will be reviewed on a yearly basis as required by FDA regulations. Periodic psychometric assessment reviews will occur at a priori defined time points to address any significant risks to quality, safety, or efficacy of the Clinical Trial, in addition to any significant risks to human subjects.

#### 4. APPLICABLE REGULATIONS AND GUIDELINES

| 21 CFR 812.40 | General Responsibilities of NRX |
|----------------|----------------------------------------------------|
| 21 CFR 812.43 | Selecting Investigators and Monitors |
| ICH E6, 2.8 | The Principles of ICH GCP |
| ICH E6, 5.5 | Trial Management, Data Handling and Record Keeping |
| ICH E6, 5.18.2 | Selection and Qualification of Monitors |

# 5. REFERENCES TO OTHER APPLICABLE SOPS & SOURCE DOCUMENTATION This SOP affects all other SOPs.

#### 6. ATTACHMENTS

GA 103-A: NRX Rater Training Guidelines [V4]

**GA 103-B: Rater Experience Survey** 

GA 103-C: NRX 101-003 Psychometric Rater Training 22Aug22 V5

GA 104-D: Rater Qualification Approval Form

#### 7. PROCESS OVERVIEW

General Training and Documentation Plan is defined in: GA 103-C: NRX 101-003 Psychometric Rater Training 22Aug22\_V5

- 1. General Training
- 2. Protocol-Specific Training
- 3. Training Documentation filed in accordance with Institutional and FDA Regulations
- 4. Periodic Review & Retraining (\*if necessary)

# 8. SPECIFIC PROCEDURES

# A. Training Plan

# 1. Initial Training

| # | Who | Task | Attachment | Related<br>SOP |
|---|---|---|---|---|
| 1. | < <nrx manager="" program="" rater="">&gt;</nrx> | Provide an appropriate period of time for Psychometricians to demonstrate understanding of General & Study-specific requirements, typically 14 days from SIV. | | |
| 2. | < <nrx manager="" program="" rater="">&gt;</nrx> | Supervise all Rater training and ensure validity and reliability of psychometric assessments following GA-103C | GA 103-C:<br>Psychometric<br>Rater<br>Training | |
| | Notes: | | | |

# 2. Continuing Education

| # | Who | Task | Attachment | Related<br>SOP |
|---|---|---|---|---|
| 1. | < <nrx manager="" program="" rater="">&gt;</nrx> | Schedule additional Rater Training if psychometric validity and reliability does not occur, following GA-103C | GA 103-C:<br>Psychometric<br>Rater<br>Training | |
| | Notes: | | | |

# 3. Periodic Rater Review & Retraining

| # | Who | Task | Attachment | Related<br>SOP |
|---|---|---|---|---|
| 1. | < <nrx manager="" program="" rater="">&gt;</nrx> | Annually, review all Psychometricans to assess competence in performing clinical research related duties | | |
| 2. | < <nrx manager="" program="" rater="">&gt;</nrx> | If performance deficiencies are noted, retrain if necessary | | |
| | Notes: | | | |

# 4. Documentation of Rater Training

| # | Who | Task | Attachment | Related<br>SOP |
|---|---|---|---|---|
| 1. | < <nrx manager="" program="" rater="">&gt;</nrx> | Provide Rater Training to ensure training and experience to conduct protocolspecific assessments. | | |
| 2. | < <nrx rater<br="">Program<br/>Manager&gt;&gt;</nrx> | Maintain updated Rater training records. Provide copies of certificates of completion of external training programs to the training files and monitor employee training and compliance with annual performance evaluations. If deficiencies are identified, retrain as necessary. | GA 103-B: Rater Experience Survey & GA 104-D: Rater Qualification Approval Form | |
| | Notes: | | | |

Revision History:

| Revision | Date | Description of changes | Requested By |
|---|---|---|---|
| 1.0 | 17-Sept-2017 | Initial Release | Margaret Mitchell |
| 2.0 | 27-Feb-2023 | Reference to new Training Documents | Marc Korczykowski |

Rater Training SOP Review and Authorization:

Marc Korczykowski, MB, MA
Director Clinical Operations, Psychometrics

**Appendix 4** Medications Indicated for Use in Bipolar Disorder

| Brand Name | Generic Name |
|---|---|
| Abilify | Aripiprazole |
| Zyprexa | Olanzapine |
| Seroquel | Quetiapine |
| Risperdal | Risperidone |
| Rexulti | Brexpiprazole |
| ☐ Vraylar | Cariprazine |
| Caplyta | Lumaterperone |
| Lurasidone | Latuda |
| Ziprasidone | Geodon |
| Saphris | Asenapine |
| Eskalith, Lithobid | Lithium |
| Lamotrigine | Lamictal |
| Eprontia, Qudexy XR Sprinkle, Topamax, Topamax Sprinkle, Trokendi XR, Topiragen, Topiramate ER (Eqv-Qudexy XR) | Topiramate |
| Depakote | Divalproex sodium |
| Tegretol | Carbamazepine |
| Trileptal | Oxcarbazepine |